Official Title: Phase III, Randomized, Multicenter Double-Blind, Double Dummy

Study to Evaluate the Efficacy and Safety of Etrolizumab Compared With Infliximab in Patients With Moderate to Severe Active Ulcerative

Colitis Who Are Naive to TNF Inhibitors

NCT Number: NCT02136069

**Document Dates:** SAP Amendment Version 3: 04-May-2020

#### STATISTICAL ANALYSIS PLAN

TITLE: PHASE III, RANDOMIZED, MULTICENTER,

DOUBLE-BLIND, DOUBLÉ-DUMMY STUDY TO EVALUATE

THE EFFICACY AND SAFETY OF ETROLIZUMAB COMPARED WITH INFLIXIMAB IN PATIENTS WITH MODERATE TO SEVERE ACTIVE ULCERATIVE COLITIS

WHO ARE NAIVE TO THE INHIBITORS

**PROTOCOL NUMBER:** GA29103 (Gardenia)

STUDY DRUG: Etrolizumab

VERSION NUMBER: 3

**IND NUMBER:** 100366

**EUDRACT NUMBER:** 2013-004282-14

**SPONSOR:** F. Hoffmann-La Roche Ltd.

PLAN PREPARED BY: M.Sc.

M.Sc.

**DATE FINAL:** Version 1: 15 May 2019

**DATE AMENDED:** Version 2: 17 December 2019

Version 3: See electronic date stamp below

#### STATISTICAL ANALYSIS PLAN AMENDMENT APPROVAL

Date and Time(UTC) Reason for Signing Name

04-May-2020 14:26:34 Company Signatory

#### **CONFIDENTIAL**

This is an F. Hoffmann-La Roche Ltd document that contains confidential information. Nothing herein is to be disclosed without written consent from F. Hoffmann-La Roche Ltd.

# STATISTICAL ANALYSIS PLAN AMENDMENT RATIONALE FOR VERSION 3

- Changes to Section 4.4 (Efficacy Analysis) were made to update the methodology for handling of treatment discontinuation intercurrent events to be set to missing for continuous endpoints and remove single imputation of worst observation carried forward.
- Changes to Section 4.4.4 (Sensitivity Analyses) to add additional sensitivity analyses for key secondary endpoints as applicable.
- Changes to Appendix 4 (Per Protocol Population [Exclusion Criteria]) were made to update the list of protocol deviations specified for exclusion from the per protocol population.

Additional minor changes have been made to improve clarity and consistency.

#### **TABLE OF CONTENTS**

| ST | | ANALYSIS PLAN AMENDMENT RATIONALE FOR 3 | 2 |
|----|-----------|-------------------------------------------------------|----|
| 1. | BACKGRO | DUND | 7 |
| 2. | STUDY DE | ESIGN | 7 |
| | 2.1 | Protocol Synopsis | 8 |
| | 2.2 | Outcome Measures | 8 |
| | 2.3 | Determination of Sample Size | 9 |
| | 2.3.1 | Sample Size | 9 |
| | 2.4 | Analysis Timing | 9 |
| 3. | STUDY CO | ONDUCT | 9 |
| | 3.1 | Randomization | 9 |
| | 3.2 | Independent Review Facility | 10 |
| | 3.3 | Data Monitoring | 10 |
| 4. | STATISTIC | CAL METHODS | 10 |
| | 4.1 | Analysis Populations | 10 |
| | 4.1.1 | Modified Intent-to-Treat (mITT) Population | 10 |
| | 4.1.2 | Per Protocol Population | 10 |
| | 4.1.3 | Safety Population | 10 |
| | 4.1.4 | Pharmacokinetic (PK)-Evaluable Population | 10 |
| | 4.2 | Analysis of Study Conduct | 10 |
| | 4.3 | Analysis of Treatment Group Comparability | 11 |
| | 4.4 | Efficacy Analysis | 11 |
| | 4.4.1 | Primary Efficacy | 12 |
| | 4.4.1.1 | Primary Treatment Effect | 12 |
| | 4.4.1.2 | Primary Efficacy Endpoint | 12 |
| | 4.4.1.3 | Clinical Responders and Clinical Remission Definition | 13 |
| | 4.4.2 | Secondary Efficacy Endpoints | 13 |
| | 4.4.2.1 | Control of Type I Error | 13 |
| | 4.4.2.2 | Clinical Remission | 14 |

| | 4.4.2.3 | Improvement in Endoscopic Appearance of the Mucosa | 15 |
|---|---|---|---|
| | 4.4.2.4 | Endoscopic Remission | |
| | 4.4.2.5 | Corticosteroid-Free Clinical Remission at Week 54 (Off Corticosteroid for At Least 24 Weeks Prior to Week 54) in Patients Who Were Receiving Corticosteroids at Baseline | 16 |
| | 4.4.2.6 | Clinical Remission at Week 54 Among patients with Clinical Response at Week 10 | 16 |
| | 4.4.2.7 | Clinical Response | 16 |
| | 4.4.2.8 | Inflammatory Bowel Disease Questionnaire (IBDQ) | 16 |
| | 4.4.3 | Exploratory Efficacy Endpoints | 17 |
| | 4.4.4 | Sensitivity Analyses | 17 |
| | 4.4.5 | Supplementary Analyses | 18 |
| | 4.4.6 | Subgroup Analyses | 18 |
| | 4.5 | Pharmacokinetic and Pharmacodynamic Analyses | 18 |
| | 4.6 | Safety Analyses | 18 |
| | 4.6.1 | Exposure of Study Medication | 18 |
| | 4.6.2 | Adverse Events | 18 |
| | 4.6.3 | Laboratory Data | 18 |
| | 4.6.4 | Vital Signs | 18 |
| | 4.6.5 | Concomitant Medications, | 18 |
| | 4.6.6 | Medical History | 18 |
| | 4.7 | Missing Data | 19 |
| | 4.8 | Interim Analyses | 19 |
| 5. | REFERE | NCES | 19 |
| | | LIST OF FIGURES | |
| Fig | ure 1 | Study Schema | 8 |
| _ | ure 2 | Multiple Testing Procedure for Endpoints | |

#### **LIST OF APPENDICES**

| Appendix 1 | Protocol Synopsis | 20 |
|------------|----------------------------------------------|----|
| | Schedule of Assessments | |
| Appendix 3 | Rescue Therapy | 39 |
| | Per Protocol Population (Exclusion Criteria) | |

#### **GLOSSARY OF ABBREVIATIONS**

AE adverse event

CCOD clinical cutoff date

CI confidence interval

CMH Cochran Mantel Haenszel

CS corticosteroids

ES Endoscopic Subscore

Etro etrolizumab

IBDQ Inflammatory Bowel Disease Questionnaire

ICE intercurrent event

INFX infliximab

IxRS interactive voice/web based response system

MCS Mayo Clinic Score

mITT modified intent-to-treat

mMCS modified Mayo Clinic Score

OLE open-label extension

PBO placebo

PK pharmacokinetic

pMCS partial Mayo Clinic Score

PP per protocol

SAP Statistical Analysis Plan

SM safety monitoring

TNF tumor necrosis factor

UC ulcerative colitis

#### 1. BACKGROUND

This Statistical Analysis Plan (SAP) describes the analyses to be performed for Study GA29103. Study GA29103 is part of a large Phase III development program for etrolizumab. Details which are common among Studies GA28950, GA29102, GA28948, GA28949, and GA29103 are described in the project SAP.

Study GA29103 is a treat-through induction and maintenance study; however, given the treat-through design, the study will not be reported in two distinct Induction and Maintenance Phases (in contrast to the GA28950 and GA29102 etrolizumab studies which incorporate the randomized withdrawal Maintenance Phase). Therefore patients are not required to reach clinical response criteria to be entered into the Maintenance Phase.

The study will be reported once data from the Week 54 treatment period has been collected in the database and data have been cleaned and verified. This will be referred to as the primary analysis.

#### 2. <u>STUDY DESIGN</u>

Study GA29103 is a multicenter, Phase III, double-blind, head-to-head study evaluating the safety, efficacy, and tolerability of etrolizumab compared to infliximab. The population is made up of moderate to severe ulcerative colitis (UC) patients who are naive to tumor necrosis factor (TNF) inhibitors (see Figure 1).

Figure 1 Study Schema



6-MP=6-mercaptopurine; AZA=azathioprine; CS= corticosteroid; EP=endpoint; OLE=open label extension; OLE-SM=open label extension–safety monitoring study; MTX=methotrexate; Q4W=every 4 weeks; Q8W=every 8 weeks; QD=once a day; QOD=every other day; SC=subcutaneous; SM=safety monitoring; TNF-naive=naive to tumor necrosis factor inhibitor; UC=ulcerative colitis; wk=week.

Following participation in this study, patients may be eligible to participate in an open-label extension and safety monitoring (OLE-SM) study (GA28951), which consists of two parts: Part 1 (designated OLE [open-label extension]) and Part 2 (designated SM [safety monitoring]).

#### 2.1 PROTOCOL SYNOPSIS

The Protocol Synopsis is in Appendix 1. For additional details, see the Schedule of Assessments in Appendix 2.

#### 2.2 OUTCOME MEASURES

Details of efficacy, safety, and pharmacokinetics outcome measures are included in the Protocol Synopsis (Appendix 1). Baseline throughout this document is defined as the last available assessment prior to first receipt of study drug.

#### 2.3 DETERMINATION OF SAMPLE SIZE

#### 2.3.1 Sample Size

Approximately 390 patients will be randomized in a 1:1 ratio to etrolizumab + infliximab dummy or infliximab + etrolizumab dummy. The sample size of N≈195 patients per group provides approximately 80% power to detect a clinically meaningful difference of 12% (18% vs. 30%) between the two groups for the primary endpoint of proportion of patients with clinical response at Week 10 and clinical remission at Week 54, using a two-sided test at a significance level of 0.05.

#### 2.4 ANALYSIS TIMING

The primary analysis will be conducted once the last patients visit to completed their Week 54 treatment period or discontinue from the study treatment has been conducted. The date associated with this visit will be termed the clinical cutoff date (CCOD) for the primary analysis, and data in the study database to the CCOD will be cleaned and verified. Sponsor personnel will be unblinded to treatment assignment to perform the primary analysis. Patients and study site personnel will remain blinded to individual treatment assignment until after the study is completed (after all patients have either completed the safety follow-up periods or discontinued early from the study) and the database is locked.

Additional analyses will be conducted once all patients have completed 12-week safety follow-up and the database has been locked. These analyses will report all adverse events (AEs) including the data collected in the 12-week safety follow-up period.

#### 3. STUDY CONDUCT

#### 3.1 RANDOMIZATION

Details of the randomization process are included in the project SAP, Section 3.1. The statistical analyses will be conducted using the stratification factors entered into the interactive voice/web based response system (IxRS) system at randomization. Sensitivity analysis of the primary endpoints using data collected in the clinical database will be conducted as required, if the database does not match IxRS due to incorrect stratification data being collected in IxRS at randomization. Due to low or zero counts in any one stratum, the stratification factors may need to be combined or removed in the primary analysis to ensure the Cochran-Mantel-Haenszel (CMH) test is not invalidated.

Patients were randomized at baseline to etrolizumab+infliximab dummy or infliximab+etrolizumab dummy using a 1:1 ratio and a permuted blocks stratified randomization (dynamically generated). Patients were stratified using the following stratification factors:

- Concomitant treatment with corticosteroids (CS) at baseline (yes/no)
- Concomitant treatment with immunosuppressants at baseline (yes/no)
- Disease activity at screening (Mayo Clinic Score [MCS] ≤9/MCS ≥10)

#### 3.2 INDEPENDENT REVIEW FACILITY

Details are included in the project SAP, Section 3.2.

#### 3.3 DATA MONITORING

Details are included in the project SAP, Section 3.3.

#### 4. STATISTICAL METHODS

#### 4.1 ANALYSIS POPULATIONS

#### 4.1.1 <u>Modified Intent-to-Treat (mITT) Population</u>

Efficacy analyses will be performed using a modified intent-to-treat (mITT) analysis population including all patients randomized into the study who received at least one dose of study drug with patients grouped according to the treatment assigned at randomization.

To allow consistency across the program, the mITT population is being used. This differs to terminology in the Protocol Version 7, Section 6.4, which uses intent-to-treat population. The definition of the population has not changed from what is in the protocol.

#### 4.1.2 Per Protocol Population

The per-protocol (PP) population is defined as the subset of the mITT population excluding major protocol deviations which may impact the efficacy outcome at Week 10. The list of protocol deviations leading to exclusion from the PP population can be found in Appendix 4.

#### 4.1.3 Safety Population

The safety analysis population will include all patients who received at least one dose of study drug, with patients grouped according to the treatment of the treatment arm most frequently received.

#### 4.1.4 <u>Pharmacokinetic (PK)-Evaluable Population</u>

The PK evaluable population includes patients who have received at least one dose of study drug and have at least one quantifiable concentration measured post baseline.

#### 4.2 ANALYSIS OF STUDY CONDUCT

All data available in the database up to the point the last patient has completed their Week 54 visit will be included to evaluate study conduct. This will include all available data from at the time of cutoff for the primary analysis. The following analyses will be performed to evaluate the study conduct:

- Summary of protocol deviations
- Summaries of mITT, PK-evaluable, and PP and safety populations, including numbers of patients in each population

Summary of patient disposition, including the number of doses received, the number
of patients experiencing disease worsening, reasons for patients withdrawing from
the study and from study treatment, and number of patients taking study treatment
and number of patients taking rescue therapy treatment

Disease worsening can be determined between and including Week 10 and Week 54 if there is

 An increase in the partial Mayo Clinic Score (pMCS)≥3 points from Week 10 and an absolute pMCS≥5 AND an endoscopic subscore of≥2,

OR

• absolute pMCS≥7 AND an endoscopic subscore of≥2

Details of the pMCS assessment are available in the project SAP in Section 4.4.2.1.

#### 4.3 ANALYSIS OF TREATMENT GROUP COMPARABILITY

Details are included in the project SAP, Section 4.3.

#### 4.4 EFFICACY ANALYSIS

All statistical hypotheses for the primary and key secondary endpoints will be evaluated under a multiple testing procedure to ensure an overall type I error no greater than 5%. Details on this testing procedure are provided in Section 4.4.3.

All comparisons between the etrolizumab and infliximab arms for binary data will use the CMH test statistic stratified by the IxRS stratification factors described in Section 3.1. For all analyses where comparison back to baseline is made, the baseline is defined as the last available assessment prior to first receipt of study drug.

In alignment with the addendum to ICH E9, the primary efficacy treatment effect (estimands) is described for the primary treatment effect in Section 4.1.1. The estimand attributes include the following two intercurrent events: treatment discontinuation and use of rescue medication as described below.

- Treatment discontinuation: All patients who discontinue study drug during the treatment period will not be assessed for any future efficacy time points (Week 10 and/or Week 54) past the study day they discontinued study drug. Therefore, these patients will be assumed to be non-responders within the categorical endpoint analyses. For continuous endpoints (e.g., Inflammatory Bowel Disease Questionnaire [IBDQ]), these patients' data will be set to missing. Handling of missing data is described in the project SAP, Section 4.8.
- Use of rescue therapy: Increased or new background medications compared to
  baseline for the treatment of UC is considered rescue therapy. Rescue therapy use
  is described in the protocol and also summarized in Appendix 3. All patients
  receiving permitted rescue therapy during the study will be asked to continue the
  study through endpoint assessment and safety follow-up. All patients receiving

prohibited rescue therapy during the Week 54 treatment period will be asked to enter safety follow-up, with no assessment of any future Week 10 or Week 54 endpoints. Patients who receive (permitted or prohibited) rescue medication will be considered non-responders for all time points following the time they received rescue therapy. For continuous outcomes (e.g., IBDQ) scores collected after the first use of rescue medication will have their data imputed using the worst post-baseline score from the following assessments: the last score available prior to the start date of first rescue medication and all scores available after the start date of rescue medication use.

#### 4.4.1 **Primary Efficacy**

#### 4.4.1.1 Primary Treatment Effect

The primary treatment effect (estimand) targeted is described by the following four attributes:

- a) **Population:** Adult patients with moderate to severe active UC who are naive to TNF inhibitors
- b) **Variable:** Clinical response at Week 10 and clinical remission at Week 54.
- c) Intercurrent Event (ICE):
  - Treatment discontinuation
  - Use of rescue therapy

Details of the ICE strategy are explained in Section 4.4.

d) **Population-Level Summary:** Difference in proportion of patients between etrolizumab and infliximab treatment groups.

#### 4.4.1.2 Primary Efficacy Endpoint

The primary efficacy endpoint is the difference in the proportion of patients in clinical response at Week 10 and clinical remission at Week 54 between the etrolizumab and infliximab treatment patients.

# Proportion of patients in clinical response at Week 10 and clinical remission at Week 54

 $= \frac{\text{\#of patients in clinical response at Week 10 and clinical remission at Week 54}}{\text{\# of patients in mITT}}$ 

The calculation will be done within treatment groups using the mITT population

**Null hypothesis H0:**  $\rho$  Etro- $\rho$  INFX=0; the proportion of patients achieving clinical response at Week 10 and clinical remission at Week 54 in the infliximab arm is the same as the proportion of patients achieving clinical response and clinical remission in the respective etrolizumab arm.

**Alternative hypothesis H1:**  $\rho$  Etro- $\rho$  INFX  $\neq$ 0; the proportion of patients achieving clinical response at Week 10 and clinical remission at Week 54 in the infliximab arm is not the same as the proportion of patients achieving clinical response and clinical remission in the respective etrolizumab arm.

#### 4.4.1.3 Clinical Responders and Clinical Remission Definition

Details of clinical responder and clinical remission and definition are provided in the project SAP, Section 4.4.2.1.4.

#### 4.4.2 <u>Secondary Efficacy Endpoints</u>

#### 4.4.2.1 Control of Type I Error

The primary and key secondary endpoints (Figure 2) will be evaluated in a hierarchical manner with multiplicity control via multistage gatekeeping under the truncated Holm multiple testing procedure (Dmitrienko et al. 2008). In Families 1 and 2 of key secondary endpoints, the same truncation parameter value of 0.5 will be applied; no truncation is applied in Family 3, since it is prioritized lowest in the hierarchy and imposes no gatekeeping restrictions on subsequent families. The truncation parameter and the relative effect sizes of the endpoints influence how power is balanced over the secondary endpoint families. Truncation parameter values close to 1 should generally be chosen when the effect sizes in high-priority endpoints are relatively large in order to maximize overall power. In other settings where the effect sizes might be smaller or mixed, a truncation parameter value closer to 0 could improve overall power. A parameter value strictly less than 1 in testing families that impose parallel gatekeeping (i.e., at least one endpoint is considered statistically significant after multiplicity adjustment in order to test the next family) is needed to achieve strong overall type I error control (Dmitrienko et al. 2009).

Under this multistage gatekeeping approach, multiplicity-adjusted p-values will reflect the gatekeeping restrictions depicted in Figure 2 In particular, the adjusted p-values for all key secondary endpoints in Families 1, 2, and 3 will be no smaller than the p-value for the primary endpoint. Similarly, the smallest adjusted p-value in Family 2 (3) will be no smaller than the smallest adjusted p-value in Family 1 (2). Endpoints for which the multiplicity-adjusted p-value is greater than 5%¹ will not be considered statistically significant. These endpoints and all endpoints not under multiplicity control will be considered to provide supportive information. By repeated application of Proposition 4.1 of Dmitrienko et al. (2008), this testing strategy ensures that the overall type I error is no greater than 5%.

<sup>&</sup>lt;sup>1</sup> The non-inferiority endpoint in Family 2 will be compared against 2.5%. Further details on this one-sided test and handling of both one sided and tw sided p values are deferred to Section 4.4.2.2

Figure 2 Multiple Testing Procedure for Endpoints

| Hierarchy | Endpoints |
|---|---|
| Primary | Clinical response at Week 10 and clinical remission at Week 54 |
| | ↓ Success on primary endpoint |
| Key secondary | Endoscopic improvement of the Mucosa at Week 54 |
| (Family 1) | Endoscopic remission at Week 54 |
| | Clinical remission at Week 54 |
| | ↓ Success on at least one endpoint |
| (Family 2) | <ul> <li>Corticosteroid-free (off corticosteroid for at least 24 weeks prior to<br/>Week 54) clinical remission at Week 54 in patients who were<br/>receiving corticosteroids at baseline</li> </ul> |
| | Clinical remission at Week 10 (non-Inferiority) |
| | ↓ Success on at least one endpoint |
| (Family 3) | Clinical remission at Week 54 among patients with a clinical response at Week 10 |
| | Clinical remission at Week 10 and Week 54 |

Ordering of endpoints within a family will be based on the p-value results from the hypotheses tests of the endpoints in Figure 2.

#### 4.4.2.2 Clinical Remission

Definition of clinical remission is provided in the project SAP, Section 4.4.2.1.4. The proportion of patients in clinical remission at Week 54, and both Week 10 and Week 54 will be analyzed using the same methods as the primary endpoint.

The difference in the proportion of patients in clinical remission between the two treatment groups (etrolizumab minus infliximab) at Week 10 will be assessed for non-inferiority.

**Null hypothesis H0:**  $\rho$  Etro- $\rho$  Infx $\leq$ -12.5%, etrolizumab is considered inferior to infliximab for clinical remission at Week 10 by more than 12.5%.

**Alternative hypothesis H1:**  $\rho$  Etro- $\rho$  Infx>–12.5%, etrolizumab is considered at least non-inferior to infliximab for clinical remission at Week 10.

95% confidence limits for the difference in clinical remission rates will be constructed using the stratified Newcombe confidence interval (Yan and Su 2010) with CMH weights. This is the same interval that will be evaluated in all stratified analysis of binary efficacy outcomes, including the primary endpoint. The non-inferiority margin of magnitude 12.5% is based on the ACT 1 and 2 placebo-controlled Phase III trials of infliximab in aTNF-naive moderate-to-severe UC patients (Rutgeerts et al. 2005). Pooling the infliximab 5 mg results presented in Table 3 of Rutgeerts et al. (2005), the treatment

effect of infliximab versus placebo on clinical remission at Week 8 is 26% (95% CI: 19%, 33%). Therefore the magnitude of the margin is below the 95% lower confidence limit for this treatment effect (19%) and represents approximately 50% of the effect point estimate (26%).

In order to adjust the non-inferiority assessment for multiplicity and to determine statistical significance, the above null and alternative hypotheses will be examined via the Farrington-Manning non-inferiority test (Farrington and Manning 1990). This test will be stratified following the approach described in Mehrotra (2001) and Wang et al. (2006), using CMH weights and null variance estimator. The nominal p-value for this stratified Farrington-Manning test will be multiplicity-adjusted as part of Family 2 in the multiple testing strategy described in Section 4.4.2.1. Note that this non-inferiority test is one-sided, whereas all other tests under multiplicity control are two-sided. In order to account for this, all nominal two-sided p-values will be converted to one-sided (by examining the direction of the effect of etrolizumab) and multiplicity adjustment will be applied to the resulting nominal one-sided p-values (ensuring strong control at 2.5%). Multiplicity-adjusted p-values will then be converted to back to two-sided p-values for all two-sided tests.

An additional analysis will be conducted where the analysis population used to assess non-inferiority is the PP population. This supplementary analysis will examine the lower limit of the stratified Newcombe confidence interval against the margin of –12.5%.

In the Study GA29103 Protocol Version 7, Section 6.4.2, 12.5% is quoted which is incorrect; the correct value is –12.5% as used above.

#### 4.4.2.3 Improvement in Endoscopic Appearance of the Mucosa

The proportion of patients with improvement in endoscopic appearance of the mucosa at Week 10, Week 54, and both Week 10 and Week 54 will be analyzed using the same methods as the primary endpoint. As detailed in Figure 2 (Section 4.4.2.1), the endpoints for Week 10 and both Week 10 and Week 54 are not included in the multiple testing procedure for endpoints. Definition of improvement in the appearance of the endoscopic mucosa is provided in the project SAP, Section 4.4.2.

#### 4.4.2.4 Endoscopic Remission

The proportion of patients with endoscopic remission at Week 54 will be analyzed using the same methods as the primary endpoint. Definition of endoscopic remission is provided in the project SAP, Section 4.4.2.1.4.

# 4.4.2.5 Corticosteroid-Free Clinical Remission at Week 54 (Off Corticosteroid for At Least 24 Weeks Prior to Week 54) in Patients Who Were Receiving Corticosteroids at Baseline

These analyses will only be conducted on a subgroup of patients who were receiving corticosteroids at baseline as per the data collected in electronic Case Report Form (e-CRF) database. Clinical Remission is defined in the project SAP, Section 4.4.2.1.4. Patients are defined as being off CS if they have no record of taking corticosteroids since the date which is twenty four weeks prior to Week 54. This date is defined as the Week 54 visit date –168 days.

Proportion of patients in corticosteroids free clinical remission at Week 54

(off corticosteroid for at least 24 weeks prior to Week 54)

in patients who were receiving corticosteroids at baseline

# of patients in clinical remission at Week 54 & off CS for 24 weeks prior to Week 54

# of patients receiving CS at baseline in the mITT

# 4.4.2.6 Clinical Remission at Week 54 Among patients with Clinical Response at Week 10

The proportion of patients in clinical remission at Week 54 among patients with clinical response at Week 10 will be analyzed using the same methods as the primary endpoint. The definition of clinical remission and clinical response is provided in the project SAP, Section 4.4.2.1.4.

Proportion of patients in clinical remission at Week 54 among patients with clinical response at Week 10

 $=\frac{\text{\# of patients with clinical response at Week 10 and in clinical remission at Week 54}}{\text{\# of patients with clinical response at Week 10}}$ 

#### 4.4.2.7 Clinical Response

Definition of clinical response is provided in the project SAP, Section 4.4.2.1.4. The proportion of patients in clinical response at Week 10 and both Week 10 and Week 54 will be analyzed using the same methods as the primary endpoint. As detailed in Figure 2 (Section 4.4.2.1), these endpoints are not included in the multiple testing procedure for endpoints.

#### 4.4.2.8 Inflammatory Bowel Disease Questionnaire (IBDQ)

Details of the IBDQ endpoint and the analyses are provided in the project SAP, Section 4.4.2.4. The change from baseline at Week 10, Week 30, and Week 54 in IBDQ between etrolizumab and infliximab treatment groups will be analyzed. As detailed in Figure 2 (Section 4.4.2.1), these endpoints are not included in the multiple testing procedure for endpoints.

#### 4.4.3 <u>Exploratory Efficacy Endpoints</u>

Exploratory endpoints detailed in the protocol will also be analyzed. Binary endpoints will use the same statistical methods used for the primary endpoint. Continuous endpoints will use the same statistical methods used for the change from baseline secondary endpoints.

#### 4.4.4 Sensitivity Analyses

To support the primary analyses the following sensitivity analyses will be conducted: definitions of pMCS and modified Mayo Clinic Score (mMCS) are included in the project SAP, Section 4.4.2.1.4.

- Proportion of patients in clinical response at Week 10 and clinical remission at Week 54 (clinical response and clinical remission derived using mMCS including mild friability in ES = 1)
- Proportion of patients in clinical response at Week 10 and clinical remission at Week 54 (clinical response and clinical remission derived using pMCS)
- Proportion of patients in clinical response at Week 10 and clinical remission at Week 54 (clinical response and clinical remission derived using mMCS excluding friability from ES=1)
- Proportion of patients in clinical response at Week 10 and clinical remission at Week 54 (tipping point analysis)

All key secondary endpoints included in Figure 2 which are calculated using MCS or the endoscopic subscore will be re analyzed as a sensitivity analyses using the mMCS excluding friability from ES=1 or the endoscopic subscore excluding friability from ES=1 if applicable. These analyses will be conducted on the mITT population and are listed below:

- Proportion of patients with improvement in endoscopic appearance of the mucosa at Week 54 (excluding friability from ES=1)
- Proportion of patients in clinical remission at Week 54 (clinical remission derived using mMCS excluding friability from ES = 1)
- Proportion of patients in corticosteroid-free clinical remission at Week 54 (off corticosteroid for at least 24 weeks prior to Week 54) in patients who were receiving corticosteroids at baseline (clinical remission derived using mMCS excluding friability from ES=1)
- Proportion of patients in clinical remission at Week 10 (clinical remission derived using mMCS excluding friability from ES = 1) (non-inferiority)
- Proportion of patients in clinical remission at Week 54 among patients with clinical response at Week 10 (clinical response and clinical remission derived using mMCS excluding friability from ES=1)
- Proportion of patients in clinical remission at Week 10 and Week 54 (clinical remission derived using mMCS excluding friability from ES=1)

#### 4.4.5 **Supplementary Analyses**

To support the primary analyses the following supplementary analyses will be conducted:

- Proportion of patients in clinical response at Week 10 and clinical remission at Week 54 (including data collected whilst patients received rescue therapy)
- Proportion of patients in clinical response at Week 10 and clinical remission at Week 54 (using logistic regression model).
- Proportion of patients in clinical response at Week 10 and remission at Week 54

#### 4.4.6 <u>Subgroup Analyses</u>

Subgroup analyses are detailed in the project SAP, Section 4.4.3.

#### 4.5 PHARMACOKINETIC AND PHARMACODYNAMIC ANALYSES

Details are included in the project SAP, Section 4.5.

#### 4.6 SAFETY ANALYSES

Data reported will include data for all patients in the safety population from baseline up until the patient completes/withdraws from the study. If a patient is ongoing in the study due to being in safety follow-up at the time of the primary data analyses, all available data at time of the CCOD will be reported. Baseline is defined as the last available assessment prior to first receipt of study drug.

Further details of the safety analyses are provided in the project SAP, Section 4.7.

#### 4.6.1 <u>Exposure of Study Medication</u>

The number of etrolizumab injections or infliximab vials will be summarized using descriptive statistics.

#### 4.6.2 Adverse Events

Details are included in the project SAP, Section 4.7.1.

#### 4.6.3 <u>Laboratory Data</u>

Details are included in the project SAP, Section 4.7.2.

#### 4.6.4 Vital Signs

Details are included in the project SAP, Section 4.7.3.

#### 4.6.5 Concomitant Medications,

Details are included in the project SAP, Section 4.7.5.

#### 4.6.6 Medical History

Details are provided in the project SAP, Section 4.7.4.

#### 4.7 MISSING DATA

Details are included in the project SAP, Section 4.8.

#### 4.8 INTERIM ANALYSES

No efficacy interim analyses are planned, or have been undertaken.

#### 5. REFERENCES

- Dmitrienko A, Tamhane AC, Wiens BL. General multistage gatekeeping procedures. Biom J. 2008;50(5):667–77.
- Dmitrienko A, Tamhane AC, Bretz F, editors. Multiple testing problems in pharmaceutical statistics. CRC Press 2009;165–91.
- Farrington C, Manning G. Test statistics and sample size formulae for comparative binomial trials with null hypothesis of non–zero risk difference or non–unity relative risk. Statistics in medicine. 1990;9(12):1447-54.
- Mehrotra DV. Stratification Issues with Binary Endpoints. Drug Information Journal: DIJ / Drug Information Association 2001;35(4):1343–50.
- Rutgeerts P, Sandborn WJ, Feagan BG, et al. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med 2005;353:2462–76.
- Wang WWB., Mehrotra DV, Chan ISF, Heyse JF. 2006. Statistical Considerations for NonInferiority/Equivalence Trials in Vaccine Development. Journal of Biopharmaceutical Statistics 2006;16(4):429–41.
- Yan X, Su XG. Stratified Wilson and Newcombe Confidence Intervals for Multiple Binomial Proportions. Statistics in Biopharmaceutical Research 2010;2(3):329–35.

#### **Appendix 1 Protocol Synopsis**

PHASE III, RANDOMIZED, MULTICENTER, DOUBLE-BLIND,
DOUBLE-DUMMY STUDY TO EVALUATE THE EFFICACY AND

SAFETY OF ETROLIZUMAB COMPARED WITH INFLIXIMAB IN PATIENTS WITH MODERATE TO SEVERE ACTIVE ULCERATIVE

**COLITIS WHO ARE NAIVE TO TNF INHIBITORS** 

PROTOCOL NUMBER: GA29103

**VERSION NUMBER:** 7

**EUDRACT NUMBER**: 2013-004282-14

**IND NUMBER:** 100366

**TEST PRODUCT:** Etrolizumab (PRO145223, RO5490261)

PHASE:

**INDICATION:** Ulcerative colitis

SPONSOR: F. Hoffmann-La Roche Ltd

#### **Objectives**

TITLE:

#### **Efficacy Objectives**

The primary efficacy objective for this study is as follows:

To evaluate the efficacy of etrolizumab (105 mg subcutaneous [SC] every 4 weeks [Q4W]) compared with infliximab in achieving <u>both</u> clinical response at Week 10 and clinical remission at Week 54 in patients with ulcerative colitis (UC) as determined by the Mayo Clinic Score (MCS).

Secondary efficacy objectives for this study are as follows:

- To evaluate clinical remission at Week 10
- To evaluate clinical remission at Week 54
- To evaluate clinical remission achieved at both Week 10 and Week 54
- To evaluate clinical remission at Week 54 among patients with a clinical response at Week 10
- To evaluate improvement in endoscopic appearance of the mucosa at Week 10
- To evaluate improvement in endoscopic appearance of the mucosa at Week 54
- To evaluate improvement in endoscopic appearance of the mucosa achieved at <u>both</u> Week 10 and Week 54
- To evaluate endoscopic remission at Week 54
- To evaluate clinical response at Week 10
- To evaluate clinical response achieved at <u>both</u> Week 10 and Week 54
- To evaluate corticosteroid-free clinical remission at Week 54 (off corticosteroids for at least 24 weeks prior to Week 54) in patients who were receiving corticosteroids at baseline
- To evaluate change from baseline in patient-reported health-related quality of life (QOL) at Weeks 10, 30, and 54, as assessed by the Inflammatory Bowel Disease Questionnaire (IBDQ)

The exploratory efficacy objectives for this study are as follows:

- To evaluate remission at Week 10
- To evaluate remission at Week 54
- To evaluate remission at both Week 10 and Week 54
- To evaluate change in health utilities, as assessed by the EuroQoL Five-Dimension Questionnaire (EQ-5D), from baseline to Weeks 10, 30, and 54
- To evaluate the frequency and duration of hospitalizations from baseline to Week 54

#### **Safety Objectives**

The safety objectives for this study are as follows:

- To evaluate the overall safety and tolerability of etrolizumab over a period of 54 weeks
- To evaluate the incidence and severity of infection-related adverse events
- To evaluate the incidence of malignancies
- To evaluate the incidence and severity of hypersensitivity reactions
- To evaluate the incidence and the clinical significance of anti-therapeutic antibodies (ATAs) to etrolizumab, or if necessary, infliximab

#### **Pharmacokinetic Objectives**

The pharmacokinetic (PK) objectives for this study are as follows:

- To evaluate the etrolizumab serum concentration at the time of primary endpoint evaluation and at a predose timepoint (Week 12)
- To evaluate the interindividual variability of and potential covariate effects on etrolizumab (or potentially infliximab) serum exposure

#### **Exploratory Pharmacodynamic,** *Predictive, and Prognostic* **Objectives**

The exploratory pharmacodynamics (PD), predictive, and prognostic objectives for this study are as follows:

- To evaluate the relationship between baseline colonic mucosal and/or peripheral blood biomarkers, including, but not limited to, αE integrin, and response to study treatment
- To evaluate the expression levels of biomarkers in colonic tissue and/or peripheral blood, including, but not limited to,  $\alpha E$  integrin, at baseline and during the treatment period
- To evaluate the PD effects on biomarkers in stool samples through assessments that may include, but are not limited to, analyses of the microbiota and bacterial cultures at baseline and during the treatment period

#### Study Design

#### **Description of Study**

This is a multicenter, Phase III, randomized, double-blind, double-dummy, parallel-group study to evaluate the safety, efficacy, and tolerability of etrolizumab (105 mg SC Q4W) compared with infliximab (5 mg/kg intravenous [IV] Weeks 0, 2, and 6, then every 8 weeks [Q8W]) in the treatment of moderate to severe UC.

Patients enrolled in this study may be eligible to participate in an open-label extension and safety monitoring (OLE-SM) study (GA28951), which consists of two parts: Part 1 (designated OLE [open-label extension]) and Part 2 (designated SM [safety monitoring]).

Disease activity will be measured using the MCS, which is the current outcome measure accepted by regulatory authorities for drug development in UC. The target population consists of patients with moderately to severely active UC (defined as MCS of 6–12, endoscopy subscore of  $\geq 2$ , as determined by the central reading procedure described in protocol, a rectal bleeding subscore  $\geq 1$ , and a stool frequency subscore  $\geq 1$ ) and involvement that extends a minimum of 20 cm from the anal verge.

All patients are to be naive to tumor necrosis factor (TNF) inhibitors.

Patients must have had an inadequate response, loss of response, or intolerance to prior immunosuppressant and/or corticosteroid treatment.

Patients who are on background immunosuppressant therapy (6-MP, AZA, MTX) may be enrolled if they have received a stable dose for at least 8 weeks prior to randomization (Day 1). Such patients should continue on their stable baseline doses of their background immunosuppressant therapy throughout the study unless dose reduction or discontinuation is required due to toxicity. Generally accepted criteria for discontinuation of immunosuppressants due to toxicity include, but are not limited to, acute pancreatitis, severe leukopenia, severe thrombocytopenia, or clinically significant elevations of the liver-associated enzymes from baseline, especially in the presence of an elevated total bilirubin. The ultimate decision to reduce dose or discontinue immunosuppressants due to toxicity remains at the discretion of the investigator.

Patients on oral corticosteroid therapy (prednisone at a stable dose of  $\leq$  30 mg, or equivalent) may be enrolled according to the following criteria:

- If corticosteroid therapy is ongoing or has just been initiated, the dose has to be stable for at least 4 weeks immediately prior to randomization (Day 1)
- If corticosteroids are being tapered, the dose has to be stable for 2 weeks immediately prior to randomization (Day 1)

Such patients should continue stable doses of their background corticosteroid until Week 10, at which point a corticosteroid taper will be initiated for all patients entering the Maintenance Phase.

Initiation of corticosteroid or an increase in corticosteroid dose above the patients' entry dose (up to a maximum of 30 mg/day of prednisone [or equivalent]) will not be permitted during screening. Use of budesonide will be allowed at stable doses ( $\leq 9$  mg) provided that the dose has been stable for  $\geq 4$  weeks prior to randomization (Day 1). Oral 5-aminosalicylate (5-ASA) treatment and probiotics for the treatment of UC may be continued at a stable dose as long as the dose(s) had been stable for  $\geq 4$  weeks and  $\geq 2$  weeks, respectively, prior to randomization (Day 1). Certain concomitant treatments are prohibited (see protocol for list of all prohibited concomitant treatments).

Patients must have discontinued topical treatments for UC at least 2 weeks prior to randomization (Day 1).

The study will be divided into:

- Screening period of up to 35 days (for details see protocol)
- Double-blind treatment period of 54 weeks, composed of an Induction Phase (up to Week 10) and a Maintenance Phase (Week 10 to Week 54)
- Safety follow-up period of 12 weeks.

A total of approximately 390 patients will be recruited from approximately 200 sites. Patients will be stratified by concomitant treatment with corticosteroids (including budesonide) at baseline (yes/no), concomitant treatment with immunosuppressants at baseline (yes/no), and baseline disease activity as measured during screening (MCS  $\leq$  9 vs. MCS  $\geq$  10).

Patients completing the Maintenance Phase at Week 54, patients identified as having disease worsening between Weeks 10 and 54, or patients who receive defined rescue medication(s) may enroll in Part 1 (OLE) of Study GA28951, if eligible, where they will receive open-label etrolizumab after a brief washout phase. If they do not enroll in Part 1 (OLE) of Study GA28951, they will enter the 12-week safety follow-up period of this study and will then be requested to enroll in Part 2 (SM) of Study GA28951 for 92 weeks of extended PML monitoring.

#### **Study Drug Administration**

Following screening, patients will be randomized in a 1:1 ratio to receive 105 mg etrolizumab or 5 mg/kg infliximab. The study design is double-blind, double-dummy, so all patients will receive two study treatments, either active etrolizumab + infliximab dummy or active infliximab + etrolizumab dummy. The dummy for etrolizumab will be a matched SC placebo, whereas the dummy for infliximab will be an IV saline infusion. Patients will receive either 105 mg etrolizumab or etrolizumab dummy by SC administration Q4W until Week 52. Infliximab will be administered by IV infusion at Weeks 0, 2, and 6, then Q8W until Week 46. Consequently, administration of SC study medication and IV study medication occurs at different timepoints throughout the study.

The first 2 doses of etrolizumab/etrolizumab dummy will be administered via a prefilled syringe (PFS) by a health care professional (HCP) in the clinic. The subsequent two doses will be self-administered by the patient or administered by his or her caregiver in the clinic and monitored by the HCP.

If deemed appropriate by HCP, the remaining doses of etrolizumab/etrolizumab dummy study drug, starting at Week 16, will be self-administered by the patient or administered by his or her caregiver at home Q4W (action to be taken as a result of a hypersensitivity reaction provided in the protocol). On occasions when the patient has to attend the clinic the same day as an etrolizumab/etrolizumab dummy administration, the administration of study medication by the patient or his or her caregiver will occur at home after his or her study assessments in the clinic setting. If necessary, patients or their HCPs may choose to continue administration of study medication in the clinic. The details of study medication administration are provided in the protocol.

In addition, patients will receive either infliximab (5 mg/kg IV at Weeks 0, 2, and 6, then Q8W) or infliximab dummy (saline) IV at the same timepoints, administered in the clinic setting until Week 46.

#### **Number of Patients**

A total of approximately 390 patients will be enrolled in this study from approximately 200 sites.

#### **Target Population**

**Inclusion Criteria** 

Patients must meet the following criteria for study entry:

- Able and willing to provide written informed consent
- 18–80 years of age, inclusive
- Diagnosis of UC established at least 3 months prior to randomization (Day 1) by clinical and endoscopic evidence. This diagnosis should be corroborated by histopathology conducted at any time prior to screening and documented by a histopathology report. (Note: histopathology may be performed at screening, if no prior report is readily available.)
- Moderately to severely active UC as determined by an MCS of 6–12, with an endoscopic subscore ≥ 2 as determined by the central reading procedure, a rectal bleeding subscore ≥ 1, and a stool frequency subscore ≥ 1 during the screening period (prior to randomization [Day 1]). See also the protocol for additional information regarding this time window.
- Evidence of UC extending a minimum of 20 cm from the anal verge as determined by baseline endoscopy (flexible sigmoidoscopy or colonoscopy) performed during screening, 4–16 days prior to randomization (Day 1). See also the protocol for additional information regarding this time window.
- Naive to treatment with any TNF inhibitor therapy (including TNF inhibitor biosimilars)

 Patients must have had an inadequate response, loss of response, or intolerance to prior immunosuppressant and/or corticosteroid treatment.

Inadequate response to, loss of response to, or intolerance to prior immunosuppressant treatment is defined as one or more of the following:

Persistent signs and symptoms of active disease despite a history of at least one 12-week regimen of oral AZA ( $\geq$  1.5 mg/kg) or 6-MP ( $\geq$  0.75 mg/kg) and/or MTX ( $\geq$  15 mg/week) within the previous 5 years

Persistent signs and symptoms of active disease despite a 6-TG level of  $\geq$  230 pmol/8  $\times$  108 RBCs during at least one 12-week regimen of oral AZA or 6-MP at a stable or increasing dose within the previous 5 years(or equivalent)

History of intolerance to AZA, 6-MP, or MTX (including, but not limited to, nausea/vomiting, abdominal pain, pancreatitis, LFT abnormalities, lymphopenia, *TPMT* genetic mutation, infection) within the previous 5 years

Inadequate response, loss of response, or intolerance to corticosteroid treatment is defined as one or more of the following:

<u>Steroid refractory</u>: persistent symptoms of active disease despite treatment with at least one 4-week induction regimen that included a dose of  $\geq$  30 mg prednisone (oral) daily (or equivalent) for at least 2 weeks or IV for at least 1 week within the previous 5 years

Steroid dependent: two failed attempts to taper steroids below a dose equivalent to 10 mg prednisone (oral) daily

<u>Steroid intolerant</u>: history of intolerance to corticosteroids (including, but not limited to, Cushing's syndrome, osteopenia/osteoporosis, hyperglycemia, insomnia, infection) within the previous 5 years

Any ongoing UC therapy must be at stable doses:

May be receiving oral 5-ASA compounds provided that the dose has been stable for ≥4 weeks immediately prior to randomization (Day 1)

May be receiving oral corticosteroid therapy (prednisone at a stable dose of  $\leq$  30 mg a day, or equivalent steroid)

If corticosteroid therapy is ongoing or has recently been initiated, the dose has to be stable for at least 4 weeks immediately prior to randomization (Day 1). If corticosteroids are being tapered, the dose has to be stable for at least 2 weeks immediately prior to randomization.

May be receiving budesonide therapy at a stable dose of up to 9 mg a day for  $\geq$  4 weeks prior to randomization (Day 1)

May be receiving probiotics (e.g., Culturelle, Saccharomyces boulardii), provided that the dose has been stable for  $\geq 2$  weeks immediately prior to randomization (Day 1)

May be receiving AZA, 6-MP, or MTX, provided that the dose has been stable for  $\geq 8$  weeks immediately prior to randomization (Day 1)

• For women who are not postmenopausal (at least 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use a highly effective method of contraception during the treatment period and for at least 24 weeks after the last dose of study drug

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

• For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 24 weeks after the last dose of study drug to avoid exposing the embryo to study drug. Men must refrain from donating sperm during this same period.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

 Must have received a colonoscopy within the past year or be willing to undergo a colonoscopy in lieu of a flexible sigmoidoscopy at screening. This colonoscopy must:

Confirm disease extent (defined as 1) left-sided colitis [up to the splenic flexure],

- 2) extensive colitis [beyond the splenic flexure but not involving the entire colon], and 3) pancolitis)
- Include removal of any adenomatous polyps

Document evidence of surveillance for dysplasia for all patients with left-sided colitis of > 12 years' duration and total/extensive colitis of > 8 years' duration

#### **Exclusion Criteria**

Patients who meet any of the following criteria will be excluded from study entry:

#### **Exclusion Criteria Related to Inflammatory Bowel Disease**

- Prior extensive colonic resection, subtotal or total colectomy, or planned surgery for UC
- Past or present ileostomy or colostomy
- · Diagnosis of indeterminate colitis
- Suspicion of ischemic colitis, radiation colitis, or microscopic colitis
- Diagnosis of toxic megacolon within 12 months of initial screening visit
- Any diagnosis of Crohn's disease
- Past or present fistula or abdominal abscess
- A history or current evidence of colonic mucosal dysplasia
- Patients with any stricture (stenosis) of the colon
- Patients with history or evidence of adenomatous colonic polyps that have not been removed

#### **Exclusion Criteria Related to Prior or Concomitant Therapy**

- Any prior treatment with etrolizumab or other anti-integrin agents (including natalizumab, vedolizumab, and efalizumab)
- Any prior treatment with anti-adhesion molecules (e.g., anti-MAdCAM-1)
- Any prior treatment with rituximab
- Any treatment with tofacitinib during screening
- Use of IV steroids within 30 days prior to screening with the exception of a single administration of IV steroid
- Use of agents that deplete B or T cells (e.g., alemtuzumab or visilizumab) within 12 months prior to randomization (Day 1), with the exception of AZA and 6-MP
- Use of cyclosporine, tacrolimus, sirolimus, or mycophenolate mofetil (MMF) within 4 weeks prior to randomization (Day 1)
- Chronic nonsteroidal anti-inflammatory drug (NSAID) use (Note that occasional use of NSAIDs and acetaminophen [e.g., headache, arthritis, myalgias, or menstrual cramps] and aspirin up to 325 mg daily is permitted.)

- Patients who are currently using anticoagulants including, but not limited to, warfarin, heparin, enoxaparin, dabigatran, apixaban, rivaroxaban. (Note that antiplatelet agents such as aspirin up to 325 mg daily or clopidogrel are permitted.)
- Patients who have received treatment with corticosteroid enemas/suppositories and/or topical (rectal) 5-ASA preparations within 2 weeks prior to randomization (Day 1)
- Apheresis (i.e., Adacolumn apheresis) within 2 weeks prior to randomization (Day 1)
- Received any investigational treatment including investigational vaccines within 5 half-lives
  of the investigational product or 28 days after the last dose (whichever is greater) prior to
  randomization (Day 1) of the study
- History of moderate or severe allergic or anaphylactic/anaphylactoid reactions to chimeric, human, or humanized antibodies, fusion proteins, or murine proteins or hypersensitivity to etrolizumab (active drug substance) or any of the excipients (L-histidine, L-arginine, succinic acid, polysorbate 20)
- Patients administered tube feeding, defined formula diets, or parenteral alimentation/nutrition who have not discontinued these treatments ≥3 weeks prior to randomization (Day 1)

#### **Exclusion Criteria Related to General Safety**

- Pregnant or lactating
- Lack of peripheral venous access
- Hospitalized (other than for elective reasons) during the screening period
- · Inability to comply with study protocol, in the opinion of the investigator
- Significant uncontrolled comorbidity, such as cardiac (e.g., moderate to severe heart failure New York Heart Association [NYHA] Class III/IV), pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders (excluding UC)
- Neurologic conditions or diseases that may interfere with monitoring for PML
- History of demvelinating disease
- Clinically significant abnormalities on screening neurologic examination (PML Objective Checklist)
- Clinically significant abnormalities on the screening PML Subjective Checklist
- History of alcohol, drug, or chemical abuse ≤ 6 months prior to screening
- Conditions other than UC that could require treatment with > 10 mg/day of prednisone (or equivalent) during the course of the study
- History of cancer, including hematologic malignancy, solid tumors, and carcinoma in situ, within 5 years before screening with the following exceptions:
  - Local basal or squamous cell carcinoma of the skin that has been excised and is considered cured is not exclusionary.
  - A history of chronic myelogenous leukemia, hairy cell leukemia, melanoma, renal cell carcinoma, or Kaposi sarcoma is exclusionary irrespective of the duration of time before screening.

History of a cervical smear indicating the presence of adenocarcinoma in situ (AIS), high-grade squamous intraepithelial lesions (HSIL), or cervical intraepithelial neoplasia (CIN) of Grade > 1, is exclusionary irrespective of the duration of time before screening.

#### **Exclusion Criteria Related to Infection Risk**

- Congenital or acquired immune deficiency
- Patients must undergo screening for HIV and test positive for preliminary and confirmatory tests

- Positive hepatitis C virus (HCV) antibody test result, unless the patient (1) has undetectable HCV RNA levels for > 6 months after completing a successful course of HCV anti-viral treatment and an undetectable HCV RNA at screening or (2) has a known history of HCV antibody positivity with a history of undetectable HCV RNA for > 6 months and undetectable HCV RNA at screening in the absence of history of HCV anti-viral treatment.
- Patients must undergo screening for hepatitis B virus (HBV). This includes testing for HBsAg (HBV surface antigen), anti-HBc total (HBV core antibody total), and HBV DNA (patients who test negative for these tests are eligible for this study):

Patients who test positive for surface antigen (HBsAg+) are not eligible for this study, regardless of the results of other hepatitis B tests.

Patients who test positive only for core antibody (anti-HBc+) must undergo further testing for hepatitis B DNA (HBV DNA test).

If the HBV DNA test result is positive, the patient is not eligible for this study. In the event the HBV DNA test cannot be performed, the patient is not eligible for this study.

If the HBV DNA test is negative, the patient is eligible for this study. These patients will undergo periodic monitoring for HBV DNA during the study

- Evidence of or treatment for *Clostridium difficile* (as assessed by C. difficile toxin testing) within 60 days prior to randomization (Day 1) or other intestinal pathogens (as assessed by stool culture and ova and parasite evaluation) within 30 days prior to randomization (Day 1)
- Evidence of or treatment for clinically significant cytomegalovirus (CMV) colitis (based on the investigator's judgment) within 60 days prior to randomization (Day 1). Laboratory confirmation of CMV from a colon biopsy sample is required during screening evaluation only if clinical suspicion is high and to determine the need for CMV treatment
- History of active or latent treated tuberculosis (TB) regardless of treatment history

Patients with a history of active or latent TB (based on a positive screening assay, either purified protein derivative [PPD] skin test or QuantiFERON®TB Gold test) are not eligible for this study.

Patients with a chest X-ray (posteroanterior [PA] and lateral) within 3 months of enrollment suspicious for pulmonary TB are **not** eligible for this study.

Any immunosuppressed patient with a strong suspicion of TB exposure and no prior vaccination with bacille Calmette-Guérin (BCG) should be considered at risk for having latent TB infection.

Patients at risk for TB exposure include:

Patients who have household contact with a person with active TB

Patients living in areas with high incidence of TB

Patients who frequently visit areas with high prevalence of active TB

Patients who meet these criteria should be evaluated per local practice to exclude latent TB.

- History of recurrent opportunistic infections and/or history of severe disseminated viral infections (e.g., herpes)
- Any serious opportunistic infection within the last 6 months
- Any current or recent signs or symptoms (within 4 weeks before screening and during screening) of infection, except for the following:

Minor infections (e.g., common cold) that have, in the investigator's judgment, completely resolved prior to randomization (Day 1)

Fungal infections of the nail beds

Oral or vaginal candidiasis that has resolved with or without treatment prior to randomization (Day 1)

 Any major episode of infection requiring treatment with IV antibiotics within 8 weeks prior to screening or oral antibiotics within 4 weeks prior to screening

Treatment with antibiotics as adjunctive therapy for UC in the absence of documented infection is not exclusionary.

- Received a live attenuated vaccine within 4 weeks prior to randomization (Day 1)
- History of organ transplant

#### **Exclusion Criteria Related to Laboratory Values (at Screening)**

- Serum creatinine > 2 × upper limit of normal (ULN)
- ALT <u>or</u> AST > 3 × ULN <u>or</u> alkaline phosphatase > 3 × ULN <u>or</u> total bilirubin > 2.5 × ULN (unconjugated hyperbilirubinemia that is associated with known Gilbert's syndrome is not an exclusion criterion)
- Platelet count < 100,000/μL</li>
- Hemoglobin < 8 g/dL</li>
- Absolute neutrophil count < 1500/μL</li>
- Absolute lymphocyte count < 500/μL</li>

#### Length of Study

The total length of the treatment period will be 54 weeks. Patients who have disease worsening between Weeks 10 and 54, patients who receive defined rescue treatment(s), and patients who complete 54 weeks of the study may be given the option of enrolling in the Part 1 (OLE) of Study GA28951, where they will receive open-label etrolizumab treatment.

Those who do not enroll in Part 1 (OLE) of Study GA28951 will continue to 12 weeks of safety follow-up in this protocol (without the washout phase) and then be requested to enroll in Part 2 (SM) of Study GA28951 for 92 weeks of PML monitoring.

The total length of the study is expected to last from the first patient screened to either the last patient in last safety follow-up visit in this protocol or the last patient enrolled into Study GA28951, whichever is later.

#### **End of Study**

The end of the study is defined as the last patient last safety follow-up visit in this protocol, or last patient in this protocol enrolled in Study GA28951, whichever is later.

#### **Outcome Measures**

#### **Efficacy Outcome Measures**

The efficacy outcome measures for this study are as follows:

Primary Efficacy Outcome Measure

 Both clinical response at Week 10 and clinical remission at Week 54 in patients with UC as determined by the MCS

#### **Secondary Efficacy Outcome Measures**

- Clinical remission at Week 10
- Clinical remission at Week 54
- Clinical remission achieved at <u>both</u> Week 10 and Week 54
- Clinical remission at Week 54 among patients with a clinical response at Week 10
- Improvement in endoscopic appearance of the mucosa at Week 10
- Improvement in endoscopic appearance of the mucosa at Week 54
- Improvement in endoscopic appearance of the mucosa achieved at <u>both</u> Week 10 and Week 54
- Endoscopic remission Week 54
- Clinical response at Week 10

#### Etrolizumab—F. Hoffmann-La Roche Ltd

- Clinical response achieved at <u>both</u> Week 10 and Week 54
- Corticosteroid-free clinical remission at Week 54 (off corticosteroids for at least 24 weeks prior to Week 54) in patients who were receiving corticosteroids at baseline
- Change from baseline in patient-reported health-related QOL at Weeks 10, 30, and 54 as assessed by the IBDQ

#### **Exploratory Efficacy Outcome Measures**

- Remission at Week 10
- Remission at Week 54
- Remission at both Week 10 and Week 54
- Change in health utilities, as assessed by the EQ-5D, from baseline to Weeks 10, 30, and 54
- Frequency and duration of hospitalizations from baseline to Week 54

#### **Safety Outcome Measures**

The safety outcome measures for this study are as follows:

- Incidence and severity of adverse events
- Incidence of serious adverse events
- Incidence and severity of infection-related adverse events
- · Incidence of serious infection-related adverse events
- Incidence and severity of injection-site reactions
- Incidence of adverse events leading to study drug discontinuation
- Incidence of laboratory abnormalities
- Incidence of malignancies
- Incidence of ATAs to etrolizumab, or if necessary, infliximab
- Incidence and severity of hypersensitivity reaction events

#### **Pharmacokinetic Outcome Measures**

The etrolizumab PK assessment will be performed in a subset of etrolizumab-treated patients. The PK outcome measures for this study are as follows:

- Serum concentration 2 weeks after the first dose and at steady state during the dosing period from Week 12 to Week 54
- Serum concentration at timepoints (Weeks 10, 30, and 54)

#### **Exploratory Biomarker Outcome Measures**

The exploratory biomarker outcome measures for this study are as follows:

- Relationship between remission and baseline levels of colonic tissue biomarkers and/or peripheral blood including, but not limited to, αE integrin. *These may be outcomes predictive or prognostic of response.*
- Changes in stool biomarkers, which may include, but are not limited to, those in the microbiota and bacterial cultures, during the Induction and Maintenance Phases as compared to baseline

#### **Investigational Medicinal Products**

#### **Test Product**

Etrolizumab PFS: containing SC formulation, 105 mg given as 0.7 mL of a 150-mg/mL solution will be administered by SC injection Q4W.

#### Comparator

Infliximab, 5 mg/kg IV Weeks 0, 2, and 6, then Q8W. Each infliximab vial contains 100 mg of lyophilized infliximab antibody in a 20-mL vial for IV use. An unblinded pharmacist will reconstitute and then dilute the infliximab to a dose of 5 mg/kg and a total volume of 250 mL with sterile 0.9% sodium chloride for infusion.

#### **Non-Investigational Medicinal Products**

Patients are to continue on their baseline dose of corticosteroid (including budesonide) to the end of the Induction Phase (Week 10). Tapering of corticosteroid (including budesonide) is to be attempted during the Maintenance Phase (Week 10 to Week 54).

Immunosuppressants (AZA, 6-MP, MTX) are to continue on the patient's baseline dose of immunosuppressant to the end of induction (Week 10) and then to continue on stable doses of immunosuppressants throughout the Maintenance Phase.

Probiotics and oral 5-ASA may be continued at a stable dose throughout the study.

Occasional use of NSAIDs and acetaminophen (e.g., headache, arthritis, myalgias, and menstrual cramps) and aspirin up to 325 mg daily are permitted throughout the study.

Anti-diarrheals (e.g., loperamide, diphenoxylate with atropine) for control of chronic diarrhea are permitted throughout the study.

#### **Statistical Methods**

#### **Efficacy Analyses**

The primary and secondary efficacy analyses will include all randomized patients who received at least one dose of study drug with patients grouped according to the treatment assigned at randomization (Day 1) (intent-to-treat [ITT] population). A per-protocol population will be defined in the Statistical Analysis Plan (SAP) for the purpose of testing for non-inferiority in induction of clinical remission at Week 10.

To manage the overall type I error, the testing of hypotheses will be performed sequentially. The primary endpoint will be tested first at an overall two-sided significance level of  $\alpha = 0.05$ . The testing hierarchy for the secondary endpoints will be described in the SAP.

Unless otherwise noted, analyses of efficacy outcome measures will be stratified by the stratification factors used at randomization (Day 1): baseline corticosteroids use (yes/no), baseline immunosuppressants use (yes/no), and baseline disease severity as measured during screening (MCS  $\leq$  9/MCS  $\geq$  10).

Patients who are non-evaluable for efficacy at a specific timepoint (e.g., due to missing data or early transfer to the Part 1 [OLE] of Study GA28951) will be considered non-responders for all response/remission type endpoints. In addition, initiation of an agent not allowed in combination with etrolizumab or infliximab, an immunosuppressant, oral or topical 5-ASA (up to Week 10), or corticosteroid, or increase in dose over baseline levels for treatment of worsening disease symptoms as defined in the protocol will lead to non-responder classification thereafter.

For continuous outcomes, scores after the first use of rescue medication will be imputed using the worst post-baseline score from the following assessments: the last score available prior to the start date of first rescue medication and all scores available after the start date of rescue medication use.

In addition to the analyses described in the protocol, the following analyses will be performed for the primary efficacy endpoint and key secondary efficacy endpoints. Details of these analyses will be described in the SAP:

- Sensitivity analyses to evaluate the robustness of results to the primary analysis methods (e.g., handling of dropouts)
- Subgroup analyses to evaluate the consistency of results across prespecified subgroups (e.g., based on age, sex, race/ethnicity, baseline UC medications, baseline CS dose)

#### **Determination of Sample Size**

Approximately 390 patients will be randomized in a 1:1 ratio to etrolizumab+infliximab dummy or infliximab+etrolizumab dummy. The sample size of 195 patients per group provides approximately 80% power to detect a clinically meaningful difference of 12% (18% vs 30%) between the two groups for the primary endpoint, using a two-sided  $\chi^2$  test at a significance level of 0.05.

## **Appendix 2 Schedule of Assessments**

| Assessment | , | Etroli | zuma | b/Etr | hedul<br>olizur | nab | c) | 1 | 1 | 1 | 1 | (1 | Etroliz | | | sit/Te | elepho | one C | days)<br>contac<br>y Adn | ct Sch | | | ome) | ı | 1 | 1 | 1 | ı | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | SD -35 to -1 | 0° | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 <sup>d</sup> | 20 | 22 | 24 | 26 <sup>d</sup> | 28 | 30 | 32 | 34 <sup>d</sup> | 36 | 38 | 40 | 42 <sup>d</sup> | 46 | 48 | 50 d | 52 | 54 | UV/<br>D-<br>OLE | EW<br>/<br>W<br>O |
| Informed consent | х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Review elig bility criteria | x e | х | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Demographic data | х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Pregnancy test f | х | х | | х | | х | | х | | | | | | | | | | | | | | | | | | | | | | х |
| Vital signs<br>(BP and pulse) | х | х | | х | | х | | | х | х | | х | х | х | | х | х | х | | х | х | х | | х | х | | х | х | | х |
| ECG | х | | | | | | | | | | | | | | | | | | | | | | | | | | | х | | х |
| Chest X-ray <sup>g</sup> | х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Height | | х | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Weight | | х | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Medical history | х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Physical examination h | х | | | | | | х | | | | | | х | | | | х | | | | х | | | х | | | | х | X b | х |
| PML neurologic examination <sup>i</sup> | х | | | х | | | х | | | | | | х | | | | | | | | х | | | | | | | х | x b | х |

## Appendix 2 Schedule of Assessments (cont.)

| Assessment | | Etrol | nic Vis<br>izuma<br>Admir | b/Etr | olizur | nab | c) | | | | | (1 | ≣troliz | | | sit/Te | elepho | one C | | ct Sch | | | ome) | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | SD -35 to -1 | 0° | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 <sup>d</sup> | 20 | 22 | 24 | 26 <sup>d</sup> | 28 | 30 | 32 | 34 <sup>d</sup> | 36 | 38 | 40 | 42 <sup>d</sup> | 46 | 48 | 50 <sup>d</sup> | 52 | 54 | UV/<br>D-<br>OLE | EW/<br>WO |
| Hematology | х | х | | | | | х | | | | | | х | | | | | | | | х | | | | | | | х | X b | <b>x</b> <sup>j</sup> |
| Chemistry | х | х | | | | | х | | | | | | х | | | | | | | | х | | | | | | | х | X b | x <sup>j</sup> |
| Urinalysis | х | х | | | | | | | | | | | | | | | | | | | | | | | | | | | X b | |
| TB screen k | х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| HIV test | х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Hepatitis B and C serology <sup>1</sup> | x | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Hepatitis B DNA <sup>m</sup> | х | | | | | | х | | | | | | х | | | | | | | | х | | | | | | | х | | |
| Hepatitis C RNA (Amplicor) <sup>n</sup> | х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| PK sampling (serum) o, p | | Х | Х | | | | х | х | | | | | | | | | х | | | | | | | | | | | х | X b | x <sup>j</sup> |
| Anti-therapeutic antibody sample (serum) o, p, q | | х | | x | | | х | х° | | | | | | | | | х° | | | | | | | | | | | Хr | x b | x j r |
| Plasma sample (storage for JCV antibody testing) | х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

## Appendix 2 Schedule of Assessments (cont.)

| Assessment | | Etroli | nic Vis<br>izuma<br>Admir | b/Etr | olizur | nab | c) | | | | | (1 | Etroliz | | nic Vi | isit/Te | elepho | one C | | ct Sch | | | ome) | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | SD -35 to -1 | 0° | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 <sup>d</sup> | 20 | 22 | 24 | 26 <sup>d</sup> | 28 | 30 | 32 | 34 <sup>d</sup> | 36 | 38 | 40 | 42 <sup>d</sup> | 46 | 48 | 50 <sup>d</sup> | 52 | 54 | UV/<br>D-<br>OLE | EW/<br>WO |
| MCS (includes endoscopy) t, u | x <sup>v</sup> | | | | | | х | | | | | | | | | | | | | | | | | | | | | х | X b | <b>X</b> <sup>j,</sup><br>gg |
| pMCS (excludes endoscopy) <sup>u, w</sup> | | x <sup>v</sup> | | х | | х | | х | | | | | х | | | | х | | | | х | | | х | | | | | x b | x <sup>j</sup> |
| Stool sample collection | x × | x <sup>y</sup> | | | | | x <sup>y</sup> | | | | | | | | | | x <sup>y</sup> | | | | | | | | | | | Хy | X b | x <sup>y</sup> |
| Colonic biopsy (CMV if required) | x <sup>z</sup> | | | | | | | | | | | | | | | | | | | | | | | | | | | | x b | |
| Colonic biopsy<br>(histopathological<br>confirmation of UC if<br>required) | x <sup>aa</sup> | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Colonic biopsies (formalin) | x bb | | | | | | x cc | | | | | | | | | | | | | | | | | | | | | x cc | x b, cc | x j,<br>cc, gg |
| Colonic biopsies (for qPCR) | x bb | | | | | | x cc | | | | | | | | | | | | | | | | | | | | | x cc | x b, cc | x <sup>j,</sup> cc, gg |
| Serum sample (CRP) p | | Х | | | | | х | | | | | | | | | | | | | | | | | | | | | х | X b | <b>x</b> <sup>j</sup> |
| Serum sample (future exploratory PD) o, p | | х | х | | | | х | х | | | | | | | | | х | | | | | | | | | | | х | | x |

## Appendix 2 Schedule of Assessments (cont.)

| Assessment | | Etroli | zuma | sit Sc<br>ab/Etr<br>nistrat | olizur | nab | c) | | | | | (E | Etroliz | | | sit/Te | elepho | one C | days)<br>contac<br>y Adn | ct Sch | | | ome) | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | SD -35 to -1 | 0° | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 <sup>d</sup> | 20 | 22 | 24 | 26 <sup>d</sup> | 28 | 30 | 32 | 34 <sup>d</sup> | 36 | 38 | 40 | 42 <sup>d</sup> | 46 | 48 | 50 <sup>d</sup> | 52 | 54 | UV/<br>D-<br>OLE | EW<br>/<br>W<br>O |
| Blood sample (RNA<br>Paxgene) o, p, dd | | х | х | | | | х | | | | | | | | | | х | | | | | | | | | | | х | | х |
| Whole blood (EDTA) optional <sup>p</sup> | | х | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| IBDQ ee | | х | | | | | х | | | | | | | | | | х | | | | | | | | | | | х | | |
| EQ-5D ee | | х | | | | | х | | | | | | | | | | х | | | | | | | | | | | х | | |
| Concomitant medications | x | x | х | х | х | х | х | х | х | х | х | х | x | x | x | х | х | х | х | х | x | х | х | х | х | х | х | х | х | х |
| Adverse events | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х |
| Infliximab/<br>infliximab dummy<br>administration | | х | х | | × | | | | x | | | | x | | | | × | | | | x | | | х | | | | | | |
| Etrolizumab/<br>etrolizumab dummy<br>administration | | x | | х | | х | | х | | х | | х | | х | | х | | х | | х | | х | | | х | | х | | | |
#### **Appendix 2** Schedule of Assessments (cont.)

Ab=antibody; ATA=anti-therapeutic antibody; BP=blood pressure; CMV=cytomegalovirus; CRP=C-reactive protein; D-OLE=decision to switch to OLE; ECG=electrocardiogram; EQ-5D=EuroQoL Five-Dimension Questionnaire; eCRF=electronic case report form; EW = early withdrawal; HBV=hepatitis B virus; HCV=hepatitis C virus; HIV=human immunodeficiency virus; IBDQ=Inflammatory Bowel Disease Questionnaire; JCV=John Cunningham virus; MCS=Mayo Clinic Score; PD=pharmacodynamics; PK=pharmacokinetic; pMCS=partial Mayo Clinic Score; PML=progressive multifocal leukoencephalopathy; qPCR=quantitative polymerase chain reaction; SD=screening day; TB=tuberculosis; UC=ulcerative colitis; UV=unscheduled visit; WO=washout.

#### Notes:

- Study assessments and blood draws are to be conducted prior to study drug administration
- All colonic biopsy samples will be taken during flexible sigmoidoscopy/colonoscopy procedure.
- Etrolizumab administration at home for eligible patients on Weeks: 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 (negative urine pregnancy test, preferably performed in home setting, required prior to administration)
- <sup>a</sup> All assessments must be performed after obtaining informed consent. Endoscopy is to be performed 4–16 days prior to randomization (Day 1). The total screening period is 35 days. Under no circumstances will either window be extended.
- Unscheduled visit (including decision to switch to OLE) represents a visit that is not as per schedule of assessment and is required for an adverse event or for potential disease worsening assessment. All indicated assessments are NOT performed at each unscheduled visit. Assessments would be symptom driven (e.g., only perform PML neurologic examination if patient reports symptoms suspected of PML; for disease worsening, infectious etiologies may be investigated if clinically indicated; and confirmation of disease worsening is performed by the Mayo Clinic Score assessment). Assessments corresponding to items noted in this column should be recorded on the eCRF. Refer to Table 3 for details regarding washout and timing of enrollment in Part 1 (OLE) of Study GA28951.
- <sup>c</sup> Day 1 of Week 0.
- d Telephone contact for patients performing home administration: patients requiring in-clinic drug administration throughout the study will have their study assessments conducted in clinic or via telephone call after their clinic visit at the sites' discretion.
- e Perform prior to first administration of study drug.
- f Serum test at screening for all female patients except those who are more than 1 year postmenopausal or have had a hysterectomy. Urine test at other visits; if urine test is positive, perform a confirmatory serum test. Pregnancy test will be carried out at home once patient starts etrolizumab administration at home. Patient is to report the pregnancy test via e-diary. Patients must be instructed at screening and reminded throughout the study that in case of positive pregnancy test they must stop self-administration of study drug and call the site immediately. Do not administer etrolizumab unless the serum pregnancy test result is negative. After Week 12, pregnancy tests to be performed prior to administration and preferably in home setting at Weeks 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52.
- <sup>g</sup> Not required if normal chest X–ray result within 3 months prior to screening.
- <sup>h</sup> Full physical examination required at screening; symptom-driven physical examination at all other timepoints indicated.

### **Appendix 2** Schedule of Assessments (cont.)

- PML neurologic examination consists of the PML Subjective Checklist and the PML Objective Checklist. Administer before other assessments, as per Appendix 5.
- J Not required if unscheduled visit leads to withdrawal or decision to switch to OLE (Part 1) and assessment was previously conducted at unscheduled visit.
- k The following tests are acceptable screening assays for latent TB in this study: purified protein derivative (a tuberculin skin test reaction aka Mantoux test), INF-γ based test (e.g., QuantiFERON®-TB Gold).
- Patients must undergo screening for HBV and HCV. This includes testing for HBsAG (HBV surface antigen), anti-HBc total (HBV core antibody total), and hepatitis C antibody.
- <sup>m</sup> Enrolled patients who are hepatitis B core antibody positive should have hepatitis B DNA measured at these timepoints.
- Measurement of HCV RNA with use of the Amplicor assay is required only when the patient has a known history of HCV antibody positivity with past documentation of undetectable HCV RNA, either with or without history of anti-viral treatment. Patients with newly diagnosed HCV antibody positivity are not eligible for this study, and therefore do not require measurement of HCV RNA.
- o Samples to be collected from a subset of patients (approximately 400 at designated sites) for PK (all scheduled timepoints), ATA (indicated times) and exploratory PD assessment (all scheduled timepoints). ATA samples at baseline Week 0, Week 10, and Week 54 are to be collected from all patients and all ATA samples may be used for exploratory PD and/or PK assessment.
- <sup>p</sup> Samples are to be collected prior to dose administration (blood, serum, colonic biopsies).
- <sup>q</sup> If serum sickness or a clinically significant allergic drug reaction is suspected, Sponsor should be notified and serum for the analysis of study drug level and ATAs should be drawn and sent to the central laboratory. ATA samples may also be utilized for exploratory PD assessments or assessment of drug concentrations.
- Collection of sample for ATA is required at final or early withdrawal visit, unless it coincides with first visit in Part 1 of Study GA28951 (where a sample for ATA must be collected).
- s A blood sample to test for antibodies to JCV will be taken and stored for possible later assessment of how widespread the JCV infection is in the study population. Sample testing for the presence of JCV antibodies is not helpful in predicting risk for PML or for evaluating neurologic symptoms. The sample may be tested if there is a strong belief that this information will be helpful in managing a patient's condition.
- <sup>t</sup> Endoscopy+rectal bleeding assessment+stool frequency assessment+Physician's Global Assessment. Patients who have not undergone full colonoscopy with documented results within one year prior to screening should undergo colonoscopy in lieu or sigmoidoscopy at the screening visit to allow for screening for cancer/dysplasia (yes/no). Rectal bleeding and stool frequency to be collected daily on e-diary.
- <sup>u</sup> During screening, patients must be trained on the use of the e-diary. Patients are to complete the e-diary on a daily basis for the stool frequency and rectal bleeding score (for MCS/pMCS) from first screening visit.
- Partial MCS during screening is defined as the MCS score excluding the endoscopy score. Screening endoscopy (for the MCS) is to be performed between 4–16 days prior to randomization (Day 1) (i.e., Day –16 to Day –4. For baseline measurements, the Physician's Global

### **Appendix 2** Schedule of Assessments (cont.)

Assessment will be obtained only once, on Day 1 (prior to randomization [Day 1)]), and the Physician's Global Assessment score will be used to calculate both the baseline (screening) MCS and the baseline (Day 1) pMCS.

- w Rectal bleeding assessment + stool frequency assessment + Physician's Global Assessment. Rectal bleeding and stool frequency to be collected daily on e-diary.
- <sup>x</sup> For culture and sensitivity testing; ova, parasites, and *Clostridium difficile* toxin testing.
- <sup>y</sup> Sample analyses may include, but are not limited to, analyses of fecal calprotectin, and other exploratory PD biomarkers (such as analyses of the microbiota and bacterial cultures).
- <sup>z</sup> IF REQUIRED: If there is suspicion for clinically significant CMV colitis, one biopsy sample should be obtained from the base of the ulcer to evaluate for histological presence of CMV. Analysis should be performed locally if possible, or can be sent to a central laboratory if necessary. Result must be negative for CMV prior to dosing on Day 1.
- <sup>aa</sup> IF REQUIRED: If patient does not have previously documented histopathologic confirmation of UC as defined in the inclusion criteria, one biopsy sample can be obtained from the base of the ulcer and read locally for histopathologic confirmation of UC.
- bb In addition to the optional biopsy noted in footnote "z" and "aa" above, five pairs (10 biopsy samples) will be obtained at screening (all taken from the most inflamed area of colon within 20–40 cm of anal verge [sigmoid]). These five biopsy pairs will be sent to the central laboratory for further storage or distribution. Two pairs will be placed in stabilization buffer (such as RNAlater or a similar buffer) and stored at –80°C (one pair for diagnostic qPCR and one pair for PD biomarkers qPCR). In the United Kingdom (U.K.) sites only, one of the latter pair of biopsies (two samples) will be placed in storage solution and shipped at 4°C to the U.K. laboratory. The other three pairs will be placed in formalin and then paraffin embedded; these biopsy samples will be used for exploratory PD biomarkers and/or diagnostic biomarkers. Original biopsy location and endoscopic depth should be clearly indicated.
- A total of four pairs (8 biopsy samples) will be obtained from all patients (all taken from the most inflamed area of colon within 20–40 cm of anal verge [sigmoid]). All will be sent to the central laboratory for further storage or distribution. Two pairs will be placed in a stabilization buffer (such as RNAlater or a similar buffer) and stored at –80°C for exploratory PD biomarker and/or diagnostic biomarker qPCR.
  In the U.K. sites only, one of the latter pair of biopsies (two samples) will be placed in storage solution and shipped at 4°C to the U.K. laboratory. The other two pairs will be placed in formalin and then paraffin; these biopsy samples will be used for exploratory PD biomarkers and/or diagnostic biomarkers. Original biopsy location and endoscopic depth should be clearly indicated.
- <sup>dd</sup> Paxgene blood RNA samples must be collected after all other blood and serum samples.
- ee With the exception of Week 0, the IBDQ and EQ-5D will be completed in-clinic by the patient before any other non-PRO assessments and before the patient receives any disease-status information or study drug during that visit.
- ff Where indicated, patients must be instructed to administer study drug at home within 3 days (maximum) after clinic visit.
- <sup>99</sup> For patients exiting the treatment period early for any reason, an endoscopy to document disease activity may be performed at the discretion of the investigator.

## Appendix 3 Rescue Therapy

| Type | Description |
|---|---|
| Permitted | Initiation or escalation beyond baseline dose of the following agents for the treatment of worsening UC symptoms. |
| | • Immunosuppressants (AZA, 6-MP or MTX) |
| | <ul> <li>Oral or topical 5-ASA or corticosteroid (use of topical at baseline is among the<br/>exclusion criteria; rectal is synonymous with topical)</li> </ul> |
| | Oral corticosteroid taper starts at Week 10 for patients on CS at baseline |
| Prohibited | Any use of other immunosuppressants, including: |
| | TNF inhibitors and biosimilars thereof |
| | Cyclosporine, tacrolimus, sirolimus, or MMF |
| | Anti-adhesion molecules, including natalizumab and vedolizumab |
| | <ul> <li>Other biologics, such as efalizumab, alemtuzumab, visilizumab and rituximab,<br/>anakinra, abatacept, tocilizumab.</li> </ul> |
| | <ul> <li>Other investigational agents, including vaccines (e.g., MAP or ChAdOx2 HAV,<br/>Janus kinase (JAK) inhibitors)</li> </ul> |
| | Patients receiving prohibited rescue therapy during the study should withdraw from the study and not receive further treatment including OLE |

5-ASA=5-aminosalicylic acid; 6-MP= 6-mercaptopurine; AZA=azathioprine; CS=corticosteriods; ChAdOx2 HAV=chimpanzee adenovirus Oxford 2 Hepatitis A vaccine; JAK=Janus kinase; MAP= Mycobacterium avium subspecies paratuberculosis; MMF=mycophenolate mofetil; MTX=methotrexate; OLE=open label extension; TNF=tumor necrosis factor; UC=ulcerative colitis

## **Appendix 4 Per Protocol Population (Exclusion Criteria)**

Patients will be excluded from the PP population if they are captured in the Protocol Deviation Management System (PDMS) under the following subcategories. The subcategories listed below are based on the latest Study GA29103 Protocol (Version 7.0). This is to ensure patients are excluded using the same criteria to allow for consistency in handling of patients within the PP population. For some subcategories whether a patient is excluded from the PP population is time dependent (prior to Week 10) as the analysis being conducted on the PP population is at Week 10.

| Category | Subcategory | Time Dependent |
|---|---|---|
| , . | A | |
| Exclusion criteria | Agents that deplete B or T cells within 12 months | |
| Exclusion criteria | Any diagnosis of Crohn's disease | |
| Exclusion criteria | Any investigational treatment/vaccines within 12 w (till PA v5) | |
| Exclusion criteria | Any prior treatment with anti-adhesion molecules | |
| Exclusion criteria | Any prior treatment with other anti-integrin | |
| Exclusion criteria | Any prior treatment with rituximab | |
| Exclusion criteria | Any stricture (stenosis) of the colon | |
| Exclusion criteria | Apheresis within 2 weeks prior to Day 1 | |
| Exclusion criteria | Corticosteroid enem/suppo & or topical 5 ASA < 2Wks | |
| Exclusion criteria | CS enem/suppo and or topical 5 ASA <= 2 wks | |
| Exclusion criteria | Diagnosis of indeterminate colitis | |
| Exclusion criteria | Diagnosis of toxic megacolon within 12 months | |
| Exclusion criteria | clusion criteria IV steroids use within 30 days prior to screening | |
| Exclusion criteria | cclusion criteria Microscopic colitis | |
| Exclusion criteria Past or present ileostomy or colostomy | | |
| | , | |
| Exclusion criteria Patients who are currently using anticoagulants | | |
| Exclusion criteria | Planned surgery for UC | |
| Exclusion criteria | Prior extensive colonic resection | |
| Exclusion criteria | Radiation colitis | |
| Exclusion criteria | Subtotal or total colectomy | |

## Appendix 4 Per Protocol Population (Exclusion Criteria) (cont.)

| Category | Category Subcategory | |
|---|---|---|
| Exclusion criteria | Suspicion of ischemic colitis | |
| Exclusion criteria | Tube feeding not discontinued ≥ 3 weeks | |
| Exclusion criteria | Use of Chronic nonsteroidal anti-inflammatory drug | |
| Exclusion criteria | Use of cyclosporine within 4 weeks prior to Day 1 | |
| Exclusion criteria | Use of mycophenolate mofetil (MMF) within 4 weeks | |
| Exclusion criteria | Use of sirolimus within 4 weeks prior to Day 1 | |
| Exclusion criteria | Use of tacrolimus within 4 weeks prior to Day 1 | |
| Exclusion criteria | Evidence/treatment for Clostridium within 60 days | |
| Exclusion criteria | Evidence/treatment for CMV colitis within 60d (V3) | |
| Exclusion criteria | Treatment for intestinal pathogens within 30d | |
| Exclusion criteria | Treatment with > 10 mg/day of prednisone or equal | |
| Inclusion criteria | Able and willing to provide written IC | |
| Inclusion criteria | Active UC with a rectal bleeding subscore ≥ 1 | |
| Inclusion criteria | Active UC with a stool frequency of ≥ 1 | |
| Inclusion criteria | Inclusion criteria Active UC with an endoscopic subscore ≥ 2 | |
| Inclusion criteria | clusion criteria Moderately to severely active UC with MCS 6-12 | |
| Inclusion criteria Diagnosis of UC at least 3 months prior to day1 (V7) | | |
| Inclusion criteria Diagnosis of UC not confirmed prior to day 1 | | |
| Inclusion criteria Initiated CS, Stable/oral CS $\leq$ 30 mg qd for $\geq$ 4 w | | |
| Inclusion criteria Initiated, Stable/oral CS <=30 mg qd for≥4 w | | |
| Inclusion criteria Naive to treatment with anti TNF/inhibitors therapy | | |
| Inclusion criteria Naive to treatment with TNFInhibitor therapy | | |
| Pts must had inad.Resp./LOR, or intol. to prior IS and/or corticosterois treatment | | |
| Inclusion criteria | Inclusion criteria Stable Immunosuppressant for 8 wks prior to D1 | |
| Inclusion criteria | Inclusion criteria Stable budesonide/MMX at ≤ 9 mg/day for ≥ 4 wks | |
| Inclusion criteria Stable doses of probiotics for ≥ 2 W prior to | | |
| Inclusion criteria | nclusion criteria Stable doses of oral 5 ASA compounds for ≥ 4 wks | |
| Inclusion criteria | Tapered CS, Stable/oral CS<=30 mg qd for≥2 w | |
| Medication | Error in Study Drug Administration Y | |
| Medication | on Overdose of study medication Y | |
| Medication Patient/site staff with blinding being compromised | | Y |
| Medication | Medication Received incorrect study medication/incorrect Kit | |
| Medication | Three consecutive missed doses of study drug | Y |
| Medication | Treatment with any other investigational agent | Y |
| Medication | Treatment with any prohibited therapies | Υ |

## Appendix 4 Per Protocol Population (Exclusion Criteria) (cont.)

| Category | Subcategory | Time Dependent |
|---|---|---|
| Medication | Use of anakinra and abatacept during the study | Y |
| Procedural | Colonic mucosal dysplasia but treatment not discon | Y |
| Procedural | De novo viral infection but treatment NOT discont. | Y |
| Procedural | Major UC related surgery but study treat. Not disc | Y |
| Procedural | Missing MCS at defined timepoints | Y |
| Procedural | Non-compliance with daily/home e-diary within 7 d | Y |
| Procedural | Patient Non-compliance with study protocol | Y |
| Procedural | Patients who miss one endoscopy at EP assessment | Y |
| Procedural | Reactivated serious VI BUT treatment NOT discont. (Viral Infection) | |
| Procedural | Rescreening procedures not completed | |
| Rescreening tests/procedures not completed- updates in ( PA v 4) | | |
| Procedural | Sigmoidoscopy not done at week 10 | Y |
| Procedural | Stable doses of immunosuppressants throughout the study (V3) | Y |
| Procedural | Video unreadable | Y |

#### STATISTICAL ANALYSIS PLAN

TITLE: DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER

STUDIES OF THE EFFICACY AND SAFETY OF ETROLIZUMAB DURING INDUCTION AND/OR MAINTENANCE PHASES IN PATIENTS WITH MODERATE TO SEVERE ACTIVE ULCERATIVE COLITIS WHO HAVE BEEN PREVIOUSLY EXPOSED TO TNF

INHIBITORS OR PATIENTS WHO ARE aTNF NAÏVE

PROTOCOL NUMBER(S): RO5490261 (GA28948, GA28949, GA29102,

GA29103, GA28950)

STUDY DRUG: Etrolizumab

**VERSION NUMBER:** 3

**IND NUMBER:** 100366

**EUDRACT NUMBER:** 2013-004278-88, 2013-004280-31, 2013-004279-11,

2013 004277-27, 2013-004282-14

**SPONSOR:** F. Hoffmann-La Roche Ltd.

PLAN PREPARED BY: , M.Sc.

**DATE FINAL:** Version 1: 14 May 2019

**DATE AMENDED:** Version 2: 17 December 2019

Version 3: See electronic date stamp below.

#### STATISTICAL ANALYSIS PLAN AMENDMENT APPROVAL

Date and Time(UTC) Reason for Signing Name

04-May-2020 14:40:20 Company Signatory

#### **CONFIDENTIAL**

This is an F. Hoffmann-La Roche Ltd document that contains confidential information. Nothing herein is to be disclosed without written consent from F. Hoffmann-La Roche Ltd.

## STATISTICAL ANALYSIS PLAN AMENDMENT RATIONALE FOR VERSION 3

- Changes to Section 4.3.2 (Baseline Disease Characteristics):
  - Prior tumor necrosis factor (TNF) Category updated Naive to Unknown
- Changes in Section 4.4.2.1.1 (Stool Frequency and Rectal Bleeding):
  - For analysis at baseline Mayo Clinic Score (MCS) subscores, stool frequency (SF) and rectal bleeding (RB) calculations clarified calculation when endoscopy occurred outside of window.
- Changes in Sections 4.4.2.1.2 (Endoscopy) and 4.4.2.1.4 (Outcome Measures Derived from the MCS):
  - Replaced using the terminology of overall score with the Hybrid Score (HS)
  - Add definition Endoscopic Remission (excluding friability from mild subscore 1)
  - Add definition Improvement of the endoscopic mucosa (excluding friability from mild subscore 1)
- Changes to Section 4.4.2.3 (UC-PRO):
  - PRO analysis method of analysis of covariance (ANCOVA) removed and mixed-model repeated measures (MMRM) has been added as the primary method.
  - Clarified the bowel domain score is 0-27
- Changes to Section 4.3 (Subgroups):
  - Added in anti-drug antibodies (ADA) positive Subgroups
- Changes to Section 4.7.1 (Adverse Events):
  - Added in non-treatment emergent report
  - Added rates for Studies GA28948 and GA28949
- Changes to Section 4.8 (Missing Data):
  - For continuous endpoints worst post baseline imputation has been removed for ulcerative colitis patient-reported outcome (UC-PRO) data, and observed case analysis added as a sensitivity analysis for SF/RB and Inflammatory Bowel Disease Questionnaire (IBDQ).
  - Further clarification of when non-responder imputation will be applied to categorical endpoints has been added.
  - Clarification the tipping point analyses will be conducted for all primary endpoints across all studies.

Additional minor changes have been made to improve clarity and consistency.

#### **TABLE OF CONTENTS**

| ST | | ANALYSIS PLAN AMENDMENT RATIONALE FOR 3 | 2 |
|----|-----------|----------------------------------------------|----|
| 1. | | OUND | |
| 2. | STUDY DI | ESIGN | 7 |
| ۷. | 2.1 | Protocol Synopsis | |
| | 2.1 | Outcome Measures | |
| | 2.2 | Determination of Sample Size | |
| | 2.3 | Analysis Timing | |
| 3. | | ONDUCT | |
| | 3.1 | Randomization | |
| | 3.2 | Independent Review Facility | |
| | 3.3 | Data Monitoring | 9 |
| 4. | STATISTIC | CAL METHODS | 9 |
| | 4.1 | Analysis Populations | 9 |
| | 4.2 | Analysis of Study Conduct | 9 |
| | 4.3 | Analysis of Treatment Group Comparability | 9 |
| | 4.3.1 | Demographics | 10 |
| | 4.3.2 | Baseline Disease Characteristics | 11 |
| | 4.3.3 | Baseline Disease Medications | 12 |
| | 4.4 | Efficacy Analysis | 12 |
| | 4.4.1 | Efficacy Endpoints | 12 |
| | 4.4.2 | Endpoint Definitions | 12 |
| | 4.4.2.1 | Mayo Clinic Score | 13 |
| | 4.4.2.2 | Histologic Endpoints | 17 |
| | 4.4.2.3 | UC-PRO | 17 |
| | 4.4.2.4 | Inflammatory Bowel Disease Questionnaire | 18 |
| | 4.4.3 | Subgroup Analyses | 19 |
| | 4.5 | Pharmacokinetic and Pharmacodynamic Analyses | 19 |
| | 4.6 | Biomarker Analysis | |
| | 4.7 | Safety Analyses | |

| 4.7.1 | Adverse Events | 20 |
|--------------|--------------------------------------|----|
| 4.7.2 | Laboratory Data | 22 |
| 4.7.3 | Vital Signs | 23 |
| 4.7.4 | Medical History | 23 |
| 4.7.5 | Concomitant Medications | 23 |
| 4.8 | Missing Data | 23 |
| 4.9 | Interim Analyses | 24 |
| 5. REFE | RENCES | 25 |
| | LIST OF TABLES | |
| Table 1 | Study Descriptions | 7 |
| Table 2 | Steps for Calculating SF/RB Subscore | 14 |
| Table 3 | Outcome Measures | |
| Table 4 | Histologic Endpoints | 17 |
| | LIST OF APPENDICES | |
| Appendix 1 | | |
| Appendix 2 | | |
| Appendix 3 | | |
| Appendix 5 | | |
| Appendix 6 | | 30 |
| , appendix c | Symptoms | 31 |

#### **GLOSSARY OF ABBREVIATIONS**

AE adverse event

AESIs adverse events of special interest

ALT alanine aminotransferase

ANCOVA analysis of covariance

aTNF anti-tumor necrosis factor

AST aspartate aminotransferase

CMH Cochran-Mantel-Haenszel

CRP C-reactive protein

CRF Case Report Form

CS corticosteroid

CSR Clinical Study Report

ES Endoscopic Subscore

FFPE formalin-fixed paraffin-embedded

**HS Hybrid Sigmoid** 

IBD inflammatory bowel disease

IBDQ Inflammatory Bowel Disease Questionnaire

iDCC independent Data Coordinating Center

iDMC independent Data Monitoring Committee

IS immunosuppressant

IxRS interactive voice/web based response system

LoPO list of planned outputs

MCS Mayo Clinic Score

MedDRA Medical Dictionary for Regulatory Activities

mITT modified intent to treat

mMCS modified Mayo Clinic Score

MMRM mixed-model repeated measures

NHI Nancy Histology Index

OLE open label extension

OLI open label induction

PD pharmacodynamic

PGA Physician's Global Assessment

PK pharmacokinetic

pMCS partial Mayo Clinic Score

RB rectal bleeding

RHI Robarts Histopathological Index

SAE serious adverse event

SAP Statistical Analysis Plan

SF stool frequency

SMQ standardized MedDRA query

TNF tumor necrosis factor

UC ulcerative colitis

UC-PRO/SS Ulcerative Colitis Patient-Reported Outcome Signs and Symptoms

ULN upper limit of normal

#### Etrolizumab — F. Hoffmann-La Roche Ltd

#### **GLOSSARY OF ABBREVIATIONS**

WOCF Worse Observation Carried Forward

#### 1. BACKGROUND

This etrolizumab project Statistical Analysis Plan (SAP) describes the study design and analyses that are common to the Phase III etrolizumab studies in ulcerative colitis (UC) patients detailed in Table 1. Elements of the study design and analysis unique to the individual studies will be explained in the respective study SAPs.

**Table 1 Study Descriptions** 

| Study | Study Description |
|---|---|
| GA28948 (Hibiscus I)<br>and<br>GA28949 (Hibiscus II) | Two identical placebo-controlled induction studies assessing the efficacy and safety of etrolizumab compared to adalimumab and placebo in patients with moderate to severe active ulcerative colitis who are naive to TNF inhibitors |
| GA29102 (Laurel) | Placebo-controlled, maintenance study assessing the efficacy and safety of etrolizumab in patients with moderate to severe active ulcerative colitis who are naive to TNF inhibitors |
| GA29103 (Gardenia) | Head To Head study to evaluate the efficacy and safety of etrolizumab compared with Infliximab in patients with moderate to severe active ulcerative colitis who are naive to TNF inhibitors |
| GA28950 (Hickory) | Placebo-controlled, induction and maintenance study assessing the efficacy and safety of etrolizumab in patients with moderate to severe active ulcerative colitis who have been previously exposed to TNF inhibitors |

TNF=tumor necrosis factor.

Studies GA28950 and GA29102 are made up of two phases: Induction Phase and Maintenance Phase. For the purpose of statistical analyses, the Induction and Maintenance Phases of Studies GA28950 and GA29102 will be treated as two independent studies and analyzed separately. Studies GA28948 and GA28949 are induction studies. Study GA29103 is a treat-through study design with no re-randomization into the Maintenance Phase; therefore, the Induction and Maintenance Phases will be analyzed as one study.

The analysis of data will be performed once all the data have been collected in the database for the primary analysis as described in the study SAPs.

#### 2. STUDY DESIGN

#### 2.1 PROTOCOL SYNOPSIS

For individual study Protocol Synopses and Schedules of Assessments, refer to the study SAP Appendix 1 and Appendix 2, respectively.

#### 2.2 OUTCOME MEASURES

For individual study outcome measures, refer to the study SAPs.

#### 2.3 DETERMINATION OF SAMPLE SIZE

For details of individual study sample size, refer to the study SAPs.

#### 2.4 ANALYSIS TIMING

For details of the analysis timing for individual studies, refer to the study SAPs.

#### 3. STUDY CONDUCT

#### 3.1 RANDOMIZATION

An independent interactive voice/Web-based response system (IxRS) vendor will conduct the randomization for all studies and the independent Data Coordinating Center (iDCC) will perform regular checks of the randomization scheme using unblinded data. The patient randomization list will be generated by the IxRS with use of a pre-defined randomization specification. During study conduct the randomization list will not be available to the study sites, study monitors, project statisticians, or the Sponsor's project team. The study team will remain blinded to study drug. If unblinding is necessary for patient management (in the case of a serious adverse event [SAE]), the investigator will be able to break the treatment code by contacting the IxRS. Treatment codes should not be broken except in emergency situations. If the investigator wishes to know the identity of the study drug for any other reason, he or she should contact the Medical Monitor. The investigator should document and provide an explanation for any premature unblinding (e.g., accidental unblinding, unblinding due to an SAE as per health authority reporting requirements). The Sponsor safety reporting department (independent to the study team) will unblind the identity of the study medication for all unexpected SAEs that are considered by the investigator to be related to study drug per safety reference document(s), such as the Investigator's Brochure, Core Data Sheet, and Summary of Product Characteristics (SmPC). Details of patients who are unblinded during the study will be included in the individual study Clinical Study Reports (CSRs).

After the end of randomization, the data entered into the IxRS system will be reconciled with the data entered into the clinical database. In particular, the kit assignments and stratification factors will be checked. Discrepancies between the IxRS and clinical database will be listed in the CSR and raised as protocol deviations. The statistical analyses will be conducted using IxRS stratification factors, and sensitivity analysis using clinical database data will be conducted if required.

Further details of stratification factors for each study is included in the study SAPs.

#### 3.2 INDEPENDENT REVIEW FACILITY

The efficacy measure Mayo Clinic Score (MCS) requires endoscopic subscores to be collected. Central reading of endoscopies will be performed throughout the studies by

**Etrolizumab** — F. Hoffmann-La Roche Ltd 8/Statistical Analysis Plan Project SAP

an independent review facility. Data collected at sites as video clips are read centrally by an independent gastroenterologist experienced in inflammatory bowel disease (IBD). The independent reader will be blinded to the patient's clinical activity and treatment allocation. Reads are collected and read locally and the again centrally. The adjudication is carried out in two stages:

- 1. A second central reading is performed if the local and initial central reading do not agree or the initial central reading cannot be performed.
- 2. The local and central reading results are combined in a final Mayo Endoscopy subscore using the median among readers, rounded up to the nearest integer.

Further details are available in the Independent Review Charter.

The efficacy measure of histologic remission requires independent scoring. The histologic scoring will be performed by a small pool of central readers who are blinded both to treatment arm and timepoint. The scoring database will ensure that all slides for a given patient are scored by the same reader. Slide image scores are based on formalin-fixed paraffin-embedded (FFPE) biopsies from the most inflamed region of the sigmoid colon. Scores are queried for discrepancies between Nancy Histologic Index (NHI) and Geboes results (e.g., NHI < 4, indicating no erosions/ulcerations, and Geboes subgrades 5.3 or 5.4, indicating the presence of erosions/ulcerations). Queries may lead to the same reader reassessing the relevant slide images and revising the scores as they deem necessary. Further details are available in the Image Review Charter.

#### 3.3 DATA MONITORING

An independent Data Monitoring Committee (iDMC) will monitor safety and study conduct on an ongoing basis for all studies. The iDMC will meet approximately every 6 months. Further details are available in the iDMC Charter.

#### 4. <u>STATISTICAL METHODS</u>

#### 4.1 ANALYSIS POPULATIONS

Analysis populations are reported in the individual study SAPs.

#### 4.2 ANALYSIS OF STUDY CONDUCT

For details on the analysis of study conduct, refer to the individual study SAPs.

#### 4.3 ANALYSIS OF TREATMENT GROUP COMPARABILITY

To review treatment group comparability within each study a number of variables collected at baseline will be compared across treatment groups. Baseline is defined as the last available assessment prior to first receipt of study drug.

For continuous variables, descriptive statistics including n, mean, median, SD, minimum, and maximum will be calculated. For categorical variables, number and percentage in

each category will be displayed. The units/categories to be used are indicated within the brackets and separated by commas.

Summaries by treatment group will be presented for all analysis populations.

Demographics and baseline characteristics presented for patients in the Maintenance
Phases will use the data collected from their baseline visits.

#### 4.3.1 Demographics

Demographics presented will include:

- Age at randomization (years), descriptive statistics, and number and percentage of patients in the following categories: 18-<40, ≥40-<65, ≥65</li>
- Gender, number and percentage of patients in the following categories: male, female
- Race, number and percentage of patients in the following categories:
  - American Indian or Alaskan Native
  - Asian
  - Black or African American
  - Native Hawaiian or other Pacific Islander
  - White
  - Other (includes Other, Multiple, and Unknown)

For Listings the Race Category Other, multiple and unknown will be reported. For summaries and subgroups the combined category 'Other' will be used.

- Region, number and percentage of patients in the following categories:
  - Central /Eastern Europe
  - USA
  - Western/Northern Europe, Canada, Australia, New Zealand
  - Asia
  - Latin America
  - Other
- Ethnicity, number and percentage of patients in the following categories: Hispanic or Latino, Not Hispanic or Latino, Not reported, Unknown
- Body Weight (kg), descriptive statistics
- Body Mass Index (BMI; kg/m²), descriptive statistics
- Tobacco Use, number and percentage of patients in the following categories: Never, Previous, Current

#### 4.3.2 <u>Baseline Disease Characteristics</u>

Details of efficacy parameters definitions listed below are provided in Section 4.4.2.

- Duration of disease (years), descriptive statistics, and number and percentage of patients in the following categories:  $<3, \ge 3-<8, \ge 8$
- Disease extent, number and percentage of patients in the following categories: Left-sided colitis, Extensive colitis, Pancolitis
- Serum C-reactive protein (CRP) (mg/L), descriptive statistics, and number and percentage of patients in the following categories: ≤2.87, >2.87-≤10, >10
- Fecal calprotectin (µg/g), descriptive statistics including median, 25th and 75th percentiles and number and percentage of patients in the following categories:
   <250, ≥250-<500, ≥500</li>
- Mayo Clinic Score (MCS), descriptive statistics, and number and percentage of patients in the following categories: MCS ≤ 9, MCS ≥ 10
- Partial Mayo Clinic Score (pMCS) –Descriptive statistics
- Modified Mayo Clinic Score (mMCS) –Descriptive statistics
- Modified Mayo Clinic Score (mMCS) (excluding friability from Mayo ES=1) Descriptive statistics
- Stratification Factor MCS Score per IxRS, number and percentage of patients in each category: MCS ≤ 9, MCS ≥ 10
- Stool Frequency (SF) Descriptive statistics.
- Rectal Bleeding (RB) Descriptive statistics.
- Physician's Global Assessment (PGA) Descriptive statistics
- Endoscopy (ES) Descriptive statistics.
- Ulcerative Colitis Patient-Reported Outcomes, Signs and Symptoms (UC-PRO/SS):
   Functional Descriptive statistics
- UC-PRO/SS: Bowel Descriptive statistics
- UC-PRO: Systemic Symptoms Descriptive Statistics
- Inflammatory Bowel Disease Questionnaire (IBDQ) Descriptive statistics
- Nancy Histological Index (NHI) Descriptive statistics and frequencies (number and percentage per grade)
- Robarts Histopathological Index (RHI) Descriptive statistics and frequencies (number and percentage per grade)
- Geboes Grading Scale Score Descriptive statistics and frequencies (number and percentage per grade)

#### 4.3.3 Baseline Disease Medications

All data types are categorical and the number and percentage of patients will be presented for each category denoted in brackets.

- Corticosteroid (CS) use at baseline (yes, no)
- Stratification Factors (IxRS): Corticosteroid (CS) use at baseline (yes, no)
- Immunosuppressant (IS) use at baseline (yes, no)
- Stratification Factors (IxRS): Immunosuppressant (IS) use at baseline number (yes, no)
- Corticosteroid and Immunosuppressant categories (CS alone, IS alone, CS and IS, None)
- Prior anti-tumor necrosis factor (aTNF) medication (yes, no)
- Prior aTNF medication (1 failure, ≥2 failures, Refractory =Primary Non-response, Loss of response =Secondary Loss of Response, Intolerant, Unknown)

Prior aTNF use is only relevant for Study GA28950; all patients in other studies are aTNF-naive.

#### 4.4 EFFICACY ANALYSIS

The hierarchical priority of key secondary endpoints and analysis populations are available in the study SAPs. All formal statistical comparisons for binary data will use the Cochran-Mantel-Haenszel (CMH) test statistics stratified by the factors used at randomization as described in the study SAPs. For all analyses in both the Induction and Maintenance Phases where comparisons back to baseline are made, baseline is defined as the last available assessment prior to first receipt of study drug in the Induction Phase. For all analyses the point estimate, 95% CIs and p-value will be reported.

#### 4.4.1 Efficacy Endpoints

All primary endpoints for the studies are derived from the MCS. Further details of the individual primary endpoint evaluation and treatment effects (estimands) are provided in the study SAPs. All primary endpoints are categorical and formal statistical comparisons between the treatment arms will use the CMH test statistics stratified by the factors used at randomization. In addition, a selection of secondary endpoints across the studies evaluating remission, clinical remission and clinical response are also derived using the full MCS.

#### 4.4.2 Endpoint Definitions

This section provides endpoint definitions for endpoints common across studies. Further study specific details including analysis timepoints and populations will be included in the study SAPs.

#### 4.4.2.1 Mayo Clinic Score

The MCS is a composite endpoint made up of four components. The score ranges from 0 to 12 with higher scores indicating more severe disease.

The MCS is used to determine a number of efficacy endpoints as described in Table 3.

MCS=Stool Frequency subscore+Rectal Bleeding subscore+Endoscopy subscore+PGA subscore

#### 4.4.2.1.1 Stool Frequency and Rectal Bleeding

Stool frequency (SF) and rectal bleeding (RB) data are collected daily via patient's diaries and each day a patient provides a score between 0-3 for each component.

#### Stool Frequency Subscore 0-3

- 0 = Normal number of stools for this patient
- 1=1 to 2 stools more than normal
- 2=3 to 4 more stools than normal
- 3=5 or more stools than normal

#### Rectal Bleeding Subscore 0–3

- 0=No blood in stool
- 1=Streaks of blood with stool less than half the time
- 2=Obvious blood with stool most of the time
- 3=Blood alone passed
- Stool Frequency (SF) subscore = Average of 3 days daily diary scores
- Rectal Bleeding (RB) subscore=Worst value of 3 days daily diary scores

Table 2 summarizes the different scenarios for calculating SF/RB sub score in the analyses. The three days of daily diary data used to calculate the subscores described above are selected from the days most recent to, (but not including) a pre specified date, and this is called the 'anchor date'.

Table 2 Steps for Calculating SF/RB Subscore

| Timepoint | Scenarios to calculate SF/RB Subscore |
|---|---|
| Baseline | Scenario 1 Bowel preparation date (prior to an endoscopy) is assigned as the 'anchor' date. Three days daily diary data collected from patient's e-diary between Day -22 and the day prior to the anchor date will be selected to calculate SF/RB scores. Daily dairy days selected closest to the anchor date will be selected first |
| | Scenario 2 Bowel preparation date (prior to an endoscopy) is assigned as the 'anchor' date. If fewer than three days of daily diary data are available between Day –22 through to the day prior to the anchor date, then additional daily diary data collected post endoscopy starting with the score recorded 2 days after the endoscopy but prior to the randomization/enrollment will be selected to calculate SF/RB scores. Examples of this scenario are illustrated (see Appendix 3). |
| | Scenario 3 Randomization/Enrollment Date is assigned as the 'anchor' date, if endoscopy did not occur between Day -21 and day prior to randomization/enrollment date. Three days worth of diary data prior to the 'anchor' date will be selected to calculate SF/RB scores. Daily dairy days selected closest to the anchor date will be selected first |
| Post<br>Baseline | Scenario 1 Bowel preparation date (prior to an endoscopy) occurring within 7 days prior to the visit date is assigned as the 'anchor' date. Three daily diary days collected within the 7 days prior to post baseline visit date will be selected, to calculate SF/RB scores. Daily dairy days selected closest to the anchor date will be selected first. Visit date is the day the PGA assessment is collected. Scenario 2 |
| | Bowel preparation date (prior to an endoscopy) is assigned as the 'anchor' date. Three daily diary days collected within the 7 days prior to post baseline visit date will be selected, to calculate SF/RB scores. Daily dairy days selected closest to the anchor date will be selected first. |
| | If further days are required, data collected +2 days after endoscopy within the 7 days prior to visit date will be used. Visit date is the day the PGA assessment is collected. |
| | Scenario 3 Visit date is assigned as the 'anchor' date. Three daily diary days collected within the 7 days prior to post baseline visit date will be selected, to calculate SF/RB scores. Daily dairy days selected closest to the anchor date will be selected first. |

SF= stool frequency; RB= rectal bleeding; PGA= Physician's Global Assessment.

The change from baseline in the SF subscore and RB subscore at Week 6 between the treatment arms will be reported for GA28950, GA28949 and GA28948 studies. This data is considered non-parametric and will be reported using RANK analysis of covariance (ANCOVAs).

#### **4.4.2.1.2 Endoscopy**

Endoscopy=Assessment of segments from 3 locations (Colon Descending, Colon Sigmoid, Rectum).

Each location is scored using the following criteria:

#### Endoscopic Subscore 0-3

- 0 = Normal or inactive disease
- 1 = Mild disease (erythema, decreased vascular pattern, mild friability)
- 2=Moderate disease (marked erythema, lack of vascular pattern, friability, erosions)
- 3=Severe disease (spontaneous bleeding, ulceration)

At baseline all segments are reviewed and scored and the worst score from the three segments is recorded as the endoscopy subscore. At baseline the endoscopy score is collected – 16 to – 4 days prior to Day 1, however for analyses purposes, any endoscopy collected prior to randomization/enrollment date will be used as the baseline endoscopy score. All assessments are performed via video and assessed by both a local reader and a central reader; adjudication process is applied if required (see Section 3.2).

Post baseline the endoscopic score is the worst score of all segments which have been assessed at baseline, if the baseline endoscopy score had Sigmoid colon score  $\leq 1$ . If at baseline the sigmoid colon score was  $\geq 2$ , the post baseline endoscopy score is the sigmoid colon score value. This methodology is called the Hybrid Sigmoid (HS) model and is used as the primary method for all analyses across all studies and throughout the project and study SAP documents the HS methodology will be used when calculating endoscopic subscore.

For mMCS (excluding friability from ES=1) the patient's endoscopic subscore will be updated from ES=1 (mild disease) to ES=2 (moderate disease) if friability is present for either central reader 1 or central reader 2 at any location. All other patients' endoscopic subscores will remain the same. For all other analyses in Table 3 using the endoscopic subscore, the definition with mild friability is considered within endoscopic subscore of 1, will be used.

#### 4.4.2.1.3 Physician's Global Assessment

The PGA will be provided by the investigator as a score of 0 to 3. The status is based on the physician's overall rating of the patient's disease activity, given endoscopy, stool frequency, rectal bleeding, abdominal pain, well-being, fecal continence, observations, and physical exam findings.

#### **Physician's Global Assessment**

- 0=Normal (Subscores are 0)
- 1 = Mild disease (Subscores are mostly 1s)
- 2=Moderate disease (Subscores are 1 to 2)
- 3=Severe disease (Subscores are 2 to 3)

#### 4.4.2.1.4 Outcome Measures Derived from the MCS

The outcome measures calculated using the MCS or a selection of components from the MCS are detailed in Table 3.

**Table 3 Outcome Measures** 

| Outcome Measure | Definition |
|---|---|
| Mayo Clinic Score (MCS) | MCS (0–12) is a composite of 4 assessments, each rated from 0–3: stool frequency, rectal bleeding, endoscopy, and PGA |
| Partial Mayo Clinic Score (pMCS) | pMCS (0–9) is a composite of 3 assessments, each rated from 0–3: stool frequency, rectal bleeding, and PGA |
| Modified Mayo Clinic Score (mMCS) | mMCS (0–9) is a composite of 3 assessments, each rated from 0–3: stool frequency, rectal bleeding, and endoscopy |
| MCS Remission | $MCS \leq 2$ with individual subscores $\leq \! 1$ and a rectal bleeding subscore of 0 |
| MCS Clinical Remission | $MCS \le 2$ with individual subscores $\le 1$ |
| MCS Clinical Response | MCS with $\geq$ 3-point decrease and 30% reduction from baseline as well as $\geq$ 1-point decrease in rectal bleeding subscore or an absolute rectal bleeding score of 0 or 1 |
| pMCS Remission | pMCS $\leq$ 2, with, rectal bleeding score of 0, PGA 0–1 and stool frequency subscore 0–1 |
| mMCS Remission<br>(excluding friability from<br>ES = 1) | mMCS $\leq$ 2, with, rectal bleeding score of 0, endoscopy 0–1 and stool frequency subscore 0–1 (Friability must be Absent for ES=1) |
| mMCS Remission (including friability in ES=1) | mMCS $\leq$ 2, with, rectal bleeding score of 0, endoscopy 0–1 and stool frequency subscore 0–1 |
| pMCS Clinical Remission | pMCS $\leq$ 2, with, rectal bleeding score of 0–1, PGA 0–1 and stool frequency subscore 0–1 |
| mMCS Clinical Remission (excluding friability from ES = 1) | mMCS $\leq$ 2, with, rectal bleeding score of 0–1, endoscopy 0–1 and stool frequency subscore 0–1 (Friability must be Absent for ES=1) |
| mMCS Clinical Remission (including friability in ES=1) | mMCS $\leq$ 2, with, rectal bleeding score of 0–1, endoscopy 0–1 and stool frequency subscore 0–1 |
| pMCS Clinical Response | A decrease in the pMCS of at least 2 points and at least 30% improvement from baseline, with an accompanying decrease in the rectal bleeding score by at least one point or an absolute rectal bleeding score of 0 or 1. |
| mMCS Clinical Response<br>(excluding friability from<br>ES=1) | A decrease in the mMCS of at least 2 points and at least 30% decrease (improvement) from baseline, with an accompanying decrease in the rectal bleeding score by at least one point or an absolute rectal bleeding score of 0 or 1. (Friability must be Absent for ES=1) |
| mMCS Clinical Response (including friability in ES=1) | A decrease in the mMCS of at least 2 points and at least 30% decrease (improvement) from baseline, with an accompanying decrease in the rectal bleeding score by at least one point or an absolute rectal bleeding score of 0 or 1. |
| Improvement in endoscopic appearance of the mucosa (including friability in ES=1) | Endoscopy subscore ≤ 1 |

| Endoscopic Remission (including friability in ES=1) | Endoscopy subscore = 0 |
|---|---|
| Improvement in endoscopic appearance of the mucosa (excluding friability from ES=1) | Endoscopy subscore $\leq 1$ (Friability must be Absent for ES = 1) |

ES= Endoscopic Subscore; PGA=Physician's Global Assessment.

Endoscopy Score=1 includes mild friability criteria unless identified in the description of an endpoint above.

#### 4.4.2.2 Histologic Endpoints

For each patient, scanned images of hematoxylin and eosin stained slides of FFPE sigmoid colon biopsies are assessed by the same pathologist from among a small pool of central readers. Details of the reading process are included in Section 3.2. Each slide image is evaluated using two histologic scoring systems: NHI (Appendix 4) and Geboes Grading Scale (Appendix 5). A third score, the RHI, is derived from selected components of Geboes Grading Scale (Appendix 5).

All histologic endpoints will be evaluated only on patients who have documented neutrophilic inflammation at baseline. Neutrophilic Inflammation will be defined using the scoring system used within the analysis. The main analysis of each histologic endpoint will be conducted on the basis of NHI scoring system, and sensitivity analyses will be conducted using RHI and Geboes Grading Scale (Table 4). This data was not collected in the GA29103 study.

**Table 4 Histologic Endpoints** 

| | | Defini | ition for each scoring system | |
|---|---|---|---|---|
| Feature or<br>Outcome | Description | NHI | RHI | Geboes Grading<br>Scale |
| | Indication of neutrophilic inflammation | NHI > 1 | RHI > 3 | Geboes 2B.1–2B.3<br>or 3.1–3.3 or 4.1–4.3<br>or 5.1–5.3 |
| Histologic remission | Resolution of neutrophilic inflammation | NHI ≤1 | RHI ≤3 and<br>Geboes 2B.0<br>and 3.0 | Geboes 2B.0 and 3.0, and 4.0, and 5.0 |

NHI=Nancy Histological Index; RHI=Robarts Histopathological Index.

#### 4.4.2.3 UC-PRO

The UC-PRO questionnaire is collected in the e-diary and completed by patients for at least 9–12 consecutive days prior to a study visit as per the Schedule of Assessments in the protocol. The UC-PRO is being reported in three domains; two domains are key endpoints and reported as UC-PRO Signs and Symptoms. This data was not collected in the GA29103 study.

#### 4.4.2.3.1 Functional and Bowel Domain

Two domain scores computed for the UC-PRO Signs and Symptoms:

- Functional Symptoms
- Bowel Movement Signs and Symptoms

There is no single total score. The questions contributing to each domain are shown in Appendix 6. The functional domain score ranges from 0–12, the bowel domain score ranges from 0–27, with a higher score indicating a worse disease state. The responder definition cutoffs for the Functional and Bowel domains will be pre-specified in the Data Analysis Plan (DAP).

The daily scores contributing to the UC-PRO/SS calculation for a visit will be selected as: most recent 7 daily scores available prior to but not including a visit. (Note: a minimum of 4 days is required.)

For each item in the questionnaire, a score will be calculated for a visit by taking the average of the most recent 7 daily scores available. The domain score for a visit will then be determined, taken as the sum of the (averaged) items for each question.

The endpoint using the UC-PRO/SS is the change from baseline at Week X in UC-PRO/SS Domain as assessed by UC-PRO/SS measure.

#### Change from Baseline at Week X

#### = Week X UCPRO/SS Domain Score - Baseline UCPRO/SS Domain Score

A MMRM (Mixed Model Repeated Measures) analysis will be performed to assess the change from baseline in UC-PRO domains at Week X and will include the fixed categorical effects of treatment, visit, study stratification factors, and treatment-by-visit interaction, and the continuous covariates of the baseline continuous UC-PRO domain and baseline UC-PRO domain-by-visit interaction. An unstructured covariance matrix will be used to model the within patient errors within the MMRM.

#### 4.4.2.3.2 Systemic Symptoms Domain

The systemic symptoms domain collected by the UC-PRO tool ranges from 0-20 with a higher score indicating a worse disease state. Details of the score are in Appendix 6. The scores are summarized using the same methodology used for functional and bowel domain in Section 4.4.2.3.1.

#### 4.4.2.4 Inflammatory Bowel Disease Questionnaire

The IBDQ is a 32-item questionnaire containing four domains: bowel symptoms (10 items), systemic symptoms (5 items), emotional function (12 items), and social function (5 items).

An overall total IBDQ score will be computed by summing the individual 32-item scores. The range for the IBDQ total score is 32–224, with higher scores denoting better health-related quality of life.

The IBDQ questionnaire is administered once per visit as per the study Schedule of Assessments, and is completed by the patient at the clinic.

The change from baseline at Week X in total IBDQ

#### Change from Baseline at Week X = Week X IBDQ - Baseline IBDQ

This is analyzed by an ANCOVA model with the factors used at randomization into the Induction/Maintenance Phases as stratification variables, and the baseline IBDQ score used as a covariate.

#### 4.4.3 Subgroup Analyses

The following subgroup analyses will be conducted on the primary endpoints for all studies. The subgroup categories are listed in Section 4.3. Study specific subgroups will be included in the study SAPs as required.

The primary endpoints will be summarized by the following subgroups using data collected in the clinical database:

- Baseline MCS
- Disease Location
- Age
- Gender
- Race
- IS use at Baseline
- CS use at Baseline
- Anti-drug antibodies (ADA) –ve/+ve (+ve transient or +ve persistent status)

Additional subgroups analysis will be conducted as appropriate.

# 4.5 PHARMACOKINETIC AND PHARMACODYNAMIC ANALYSES Pharmacokinetic Analyses

Serum concentration at various times during Induction and Maintenance Phases will be listed and summarized by descriptive summary statistics including means, geometric means, ranges, SD, and coefficients of variation.

Individual and mean concentration versus time data will be tabulated and plotted if more than 2 time points are available.

The pharmacokinetic (PK) data from each individual study may be combined with data from other etrolizumab studies to perform a population PK analysis. Population typical value of PK parameters will be estimated for the entire study population, along with estimates of intra- and inter-patient variance and an estimate of random error. Individual patient parameter estimates will be computed using the post hoc analysis procedure. Impacts of covariates on relevant PK parameters will also be evaluated. A separate prospective analysis plan will be prepared, and the population PK analysis will be presented in a separate report for all studies, this will be separate from each study CSR.

#### Pharmacodynamic Analyses

The pharmacodynamic (PD) biomarker, sMAdCAM-1 absolute concentration and percentage change from baseline values will be listed and summarized by descriptive summary statistics at each time point including but not limited to means, SD, medians, and ranges. Analyses will be split by treatment group and cohort as appropriate.

Additional exploratory PK/PD analyses or modeling may be conducted as appropriate

#### 4.6 BIOMARKER ANALYSIS

Additional biomarker strategies and analyses will be detailed in the Biomarker Analysis Plan.

#### 4.7 SAFETY ANALYSES

The safety populations include all patients who received at least one dose of study drug, and patients will be grouped according to the treatment of the treatment arm they most frequently received. In addition, data will be listed for patients who do not receive the treatment they are assigned to in the safety population at any time point. All safety parameters will be summarized and presented in tables using the safety populations defined for each study. Patients who are not randomized but who receive study drug will be included in the safety population and summarized according to the therapy actually received. The safety data will be listed and summarized at the time of the primary analyses with use of all safety data available at the primary database snapshot. Additional summaries will be run once all patients have completed safety follow-up.

#### 4.7.1 Adverse Events

Adverse events (AEs) will include all terms recorded on the AE Case Report Form (CRF) pages (except pregnancies). For each recorded AE, the term entered by the investigator describing the event (the "reported term") will be assigned a standardized term (the "preferred term") and assigned to a superclass term on the basis of the Medical Dictionary for Regulatory Activities (MedDRA) World Health Organization (WHO) dictionary of terms. All analyses of AE data will be performed using the preferred terms unless otherwise specified. For all summary tables, the AEs will be sorted by System Organ Class (in decreasing order of overall incidence) and then by preferred term (in decreasing order of overall incidence). In addition, separate summaries or listings will

be generated for SAEs, deaths, AEs leading to discontinuation of study drug, and adverse events of special interest (AESIs). In addition to summaries or listings, narratives will be provided for all deaths, SAE's, AE's leading to treatment discontinuation and pregnancies as well as for all serious infections, opportunistic infections and malignancies in the individual CSRs.

For the etrolizumab Phase III program, the AESIs (identified by the investigator using the eCRF tick box) are the following:

- Systemic hypersensitivity reactions and anaphylactic and anaphylactoid reaction.
   These will be further described using the MedDRA anaphylactic reaction SMQ (Standard MedDRA Query) algorithmic and Hypersensitivity SMQ narrow.
- Neurological signs, symptoms, and AEs that may suggest possible progressive multifocal leukoencephalopathy (PML) (see Appendices 5 and 6 of Protocol)
- Suspected transmission of an infectious agent by the study drug
- Cases of potential drug-induced liver injury that include an elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law

Specific AEs listed below will also be reported:

- Serious infections (including GI) Events occurred in the MedDRA Infections and Infestations System Organ Class (SOC) using the primary coding events
- Opportunistic infections Events occurred in the Sponsor-defined Adverse Event Group Terms
- Malignancies Events that occur in the MedDRA Malignant and Unspecified Tumours SMQ (narrow).
- Injection site reactions Events identified using the eCRF tick box indicating an Injection site reaction AND/OR events occurred in the MedDRA Injection Site Reaction High Level Term (HLT) using both primary and secondary coding.

Outputs will be summarized using the safety population split by treatment arm and cohort as appropriate.

Summaries of AEs will be generated to summarize the incidence of treatment-emergent AEs only. Treatment-emergent events are defined as any new AE reported or any worsening of an existing condition on or after the first dose of study drug. If the onset date of the AE is prior to the day of first dose, the AE will be considered treatment-emergent only if the most extreme intensity is greater than the initial intensity (i.e., the intensity for a given AE increases and its end date is on or after the date of the first dose). Non-treatment emergent AE's collected in the database will also be reported separately, for each individual CSRs.

For each treatment group, the incidence count for each AE preferred term will be defined as the number of patients reporting at least one treatment-emergent occurrence of the

event (multiple occurrences of the same AE in one patient will be counted only once). The proportion of patients with an AE will be calculated as the incidence count divided by the total number of patients in the population. Each table will also present the total number of AEs reported where multiple occurrences of the same AE in an individual are counted separately.

The rate per 100 patient years and 95% CIs will be summarized by treatment group for studies (GA28950, GA29102, GA29103, GA28948, and GA28949). Rates will be calculated for AEs, SAEs, and other AE grouping as appropriate. The rate of AEs per 100 patient years is calculated as:

All summaries and listings of AEs will be based on the induction safety population or the maintenance safety population and listed in the List of Planned Outputs (LoPO).

#### 4.7.2 <u>Laboratory Data</u>

Descriptive summaries of laboratory values at baseline and throughout the studies will be summarized by treatment arm.

Change from baseline will be analysed for the following parameters: Hematology (hemoglobin, hematocrit, platelet count, WBC count, lymphocytes, mean corpuscular volume), serum chemistries (sodium, potassium, chloride, bicarbonate, glucose, blood urea nitrogen, creatinine, calcium, total and direct bilirubin, total protein, albumin, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase), CRP, and fecal calprotectin

Proportion of patients experiencing clinically significant changes relative to baseline will be summarized by treatment arm as appropriate for the parameters listed above.

Laboratory abnormalities and the patient's worst National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grade during study will be summarized by treatment arm as appropriate for parameters listed above.

Elevated liver enzyme tests will be summarized by the following upper limit of normal (ULN) categories as these are indicators of severe liver injury

- ALT or AST >3 × ULN
- ALT or AST >3 × ULN and total bilirubin >2 × ULN as defined by Hy's law:

The number and percentage of patients with positive serum antibodies to etrolizumab (ADA) at baseline (prevalence) and post etrolizumab treatment at any time during the

study (incidence) will be tabulated by treatment arm and listed alongside the primary efficacy outcome.

All summaries and listings of laboratory data will be based on the safety populations and specified in the LoPO.

#### 4.7.3 <u>Vital Signs</u>

Vital signs will be summarized using summary statistics and change from baseline proportion of patients experiencing clinically significant changes relative to baseline will be reported if appropriate.

All summaries and listings of vital signs data will be based on safety population and specified in LoPO.

#### 4.7.4 <u>Medical History</u>

Medical history data collected in the e-CRF will be summarized using summary statistics, reporting the proportion of patients with at least one medical condition and the total number of medical conditions. The medical conditions will then be split out by type.

All summaries and listings of medical history will be based on safety population and specified in the LoPO.

#### 4.7.5 <u>Concomitant Medications</u>

Concomitant medications include any medication being used at any time from first dose of study drug through to day of study discontinuation/completion, or medication being used at any time up to the start of study treatment. The data will be summarized, and report the total number of patients taking at least one medication, and total number of medications. Summaries will also be split by medication class and preferred medication.

All summaries and listings of concomitant medications will be based on safety population and specified in the LoPO.

#### 4.8 MISSING DATA

The handling of intercurrent events explained in the individual studies will be applied before using the missing data handling approaches in this section. The handling of intercurrent events will occur in the order the intercurrent event occurs within the study.

To assess the robustness of the primary endpoint, a tipping point analysis will be conducted. The tipping point is defined as the difference in the number of missing events (i.e., remission) between the treatment groups that result in a change in the primary outcome conclusions (Yan et al. 2009). A two-dimensional plot will be produced for each primary comparison of etrolizumab (105 mg) vs. the comparator to evaluate where the tipping point lies.

The tipping point analysis will be used to assess the robustness of the primary endpoints within each study. The following groups of patients will always be considered nonremitters/non-responders within the tipping point analysis.

- Patients whose remitter/responder status can be calculated as a non-remitter/non-responder from their available sub scores, even when not all four MCS subscores are available.
- Patients who have received rescue therapy during the study.
- Patients who have discontinued study treatment early.

For all continuous endpoints, a MMRM model will be fitted to analyse UC-PRO domains assuming the data is missing at random. For missing SF/RB and IBDQ data single imputation worse observation carried forward (WOCF) post baseline will be applied to missing data, including when data is missing due to intercurrent event. An additional sensitivity analysis using observed case will be conducted, to assess the robustness of the analysis. All summary data will be reported using no imputation for missing data.

For any missing baseline data, no imputation of results data will be applied, and therefore, any endpoints requiring comparison back to baseline results will also be set to missing. To prevent a missing SF/RB subscore at baseline or post baseline which would lead to a missing MCS/mMCS/pMCS score, the anchor date used for selecting diary data to calculate RB/SF subscores can be imputed. If bowel prep date is missing, then endoscopy date can be used; if the endoscopy date is missing then the visit date can be used as the anchor date. If the PGA visit date is missing, the visit date will be imputed as Day 1+x weeks to allow RB and SF scores to be calculated.

No imputation will be applied for missing laboratory or vital signs data.

An AE with a completely missing, non-imputed start date will be assumed to be treatment-emergent, unless the AE has a complete, non-imputed end date that is prior to the date of the first dose.

All deaths will be reported, regardless of completeness of death date.

#### 4.9 INTERIM ANALYSES

No interim analyses are planned for these studies.

#### 5. <u>REFERENCES</u>

- Geboes K, Riddell R, Öst A, et al. A reproducible grading scale for histological assessment of inflammation in ulcerative colitis. Gut. 2000;47(3):404–9.
- Mosli MH, Feagan BG, Zou G, et al. Development and validation of a histological index for UC. Gut. 2017;66(1):50–8.
- Marchal-Bressenot A, Scherl A, Salleron J, et al. A practical guide to assess the Nancy Histological Index for UC. Gut. 2016;65(11):1919–20.
- Marchal-Bressenot A, Salleron J, Boulagnon-Rombi C, et al. Development and validation of the Nancy Histological Index for UC. Gut. 2017;66(1):43–9.
- Yan X, Lee S, Li N. Missing data handling methods in medical device clinical trials. J Biopharm Stat. 2009;19(6):1085–98.

## **Appendix 1 Protocol Synopsis**

| See individual study SAPs for Protocol Synopsis. |
|--------------------------------------------------|

## **Appendix 2 Schedule of Assessments**

| • • |
|--------------------------------------------------------|
| See individual study SAPs for Schedule of Assessments. |

#### **Appendix 3 Mayo Clinic Score Measurement**

#### Scenario 1: Sufficient e-Diary Data Available prior to Endoscopy at Day -16

The e-diary data from the 3 consecutive days immediately preceding the bowel preparation day (Day -17 in this scenario) are used to derive RB and SF data for MCS calculation (Day -20 to Day -18, highlighted with dashed lines in the figure). If e-diary data from these days are missing, RB/SF data from the preceding days (Day -21 or Day -22) will be used. No RB/SF data can be obtained prior to Day -22.



#### \*If RB/SF data are not available, data from the preceding day (Day -21) will be used.

#### Scenario 2: Sufficient e-Diary Data Available prior to Endoscopy at Day -4

The e-diary data from the 3 consecutive days immediately preceding the bowel preparation day {Day -5 in this scenario} are used to derive RB and SF data for MCS calculation (Day -6 to Day -8, highlighted with dashed lines in the figure). If e-diary data from these days are missing, RB/SF data from the preceding days (Days -9 to Day -22) will be used. No RB/SF data can be obtained prior to Day -22.



\*If RB/SF data are not available, data from the preceding day (Day -9) will be used.

#### Scenario 3: Insufficient e-Diary Data Available prior to Endoscopy at Day -16

Only in cases where < 3 days of e-diary data are available prior to the bowel preparation day (Day –18 to Day –22 in this scenario), supplement with e-diary data starting 2 days after the endoscopy (e.g., January 28 if the endoscopy was performed on January 26). In the figure, the days highlighted with dashed lines can be used for MCS calculation.



<sup>\*</sup>If RB/SF data are not available, data from the next day (Day -13) will be used.



#### Scenario 4: Insufficient e-Diary Data Available prior to Endoscopy at Day -4

Only in cases where there are insufficient e-diary data (< 3 days total) available prior to the bowel preparation day (Day –6 to Day –22 in this scenario) and between the endoscopy and randomization (Day –2 and Day –1), the randomization visit must be delayed by at least 1 day by extending the screening period so sufficient data can be recorded in the e-diary (Day –1 in the extended screening period in Figure B). In the schema, the days highlighted with dashed lines can be used for MCS calculation.



Endo=day of endoscopy; MCS=Mayo Clinic Score; Rand=day of randomization; RB=rectal bleeding; SF=stool frequency.

### **Appendix 4 Nancy Histological Index**

Nancy Histological Index (NHI): Scoring algorithm



Source: Adapted from Marchal-Bressenot et al. 2016, Marchal-Bressenot et al 2017.

## Appendix 5 Geboes Grading Scale and Robarts Histopathological Index

Geboes Grading Scale: Grades and Subgrades

#### **Grade 0: Structural (architectural change)**

- 0.0 No abnormality
- 0.1 Mild abnormality
- 0.2 Mild-moderate diffuse/multifocal abnormalities
- 0.3 Severe diffuse/multifocal abnormalities

#### **Grade 1: Chronic inflammatory infiltrate**

- 1.0 No increase
- 1.1 Mild but unequivocal increase
- 1.2 Moderate increase
- 1.3 Marked increase

#### Grade 2A: Eosinophils in lamina propria

2A.0 No increase

- 2A.1 Mild but unequivocal increase
- 2A.2 Moderate increase
- 2A.3 Marked increase

#### Grade 2B: Neutrophils in lamina propria

2B.0 None

- 2B.1 Mild but unequivocal increase
- 2B.2 Moderate increase
- 2B.3 Marked increase

Source: Geboes et al. 2000.

#### **Grade 3: Neutrophils in epithelium**

- 3.0 None
- 3.1 < 5% crypts involved
- 3.2 < 50% crypts involved
- 3.3 > 50% crypts involved

#### **Grade 4: Crypt destruction**

- 4.0 None
- 4.1 Probable–local excess of neutrophils in part of crypt
- 4.2 Probable-marked attenuation
- 4.3 Unequivocal crypt destruction

#### **Grade 5: Erosion or ulceration**

- 5.0 No erosion, ulceration or granulation tissue
- 5.1 Recovering epithelium + adjacent inflammation
- 5.2 Probable erosion-focally stripped
- 5.3 Unequivocal erosion
- 5.4 Ulcer or granulation tissue

## Robarts Histopathological Index (RHI): Grade-Weighted Sum of Subgrades from Geboes

RHI score (0-33) = 1 × chronic inflammatory infiltrate (0-3)

+ 2 × neutrophils in lamina propria (0-3)

+ 3 × neutrophils epithelium (0-3)

+ 5 × erosion or ulceration (0-3)

Note: Erosion or ulceration component subgrade range of 0 to 3 is obtained by scoring Geboes subgrades as follows: 5.0 = 0, 5.1 or 5.2 = 1, 5.3 = 2, and 5.4 = 3.

Source: Mosli et al. 2017.

# Appendix 6 Ulcerative Colitis Patient Reported Outcomes Signs and Symptoms

| UC-PRO/SS<br>Domain | Question | Response to<br>Question |
|---|---|---|
| Functional<br>Symptoms | In the past 24 hours, did you pass gas? | 0=No<br>1=Rarely<br>2=Sometimes<br>3=Often<br>4=Very often |
| | In the past 24 hours, did you feel pain in your belly? | 0=No<br>1=Mild<br>2=Moderate<br>3=Severe<br>4=Very Severe |
| | In the past 24 hours, did you feel bloating in your belly? | 0=No<br>1=Mild<br>2=Moderate<br>3=Severe<br>4=Very Severe |

# Appendix 6 Ulcerative Colitis Patient Reported Outcomes Signs and Symptoms (contd.)

| UC-PRO/SS<br>Domain | Question | Response to<br>Question |
|---|---|---|
| Bowel Movement<br>Signs and<br>Symptoms | In the past 24 hours, how many bowel movements did you have? | 0=0,<br>1=1-2,<br>2=3-4,<br>3=5-6,<br>4=7-9,<br>5=10-12,<br>6=13-17,<br>7=18 or more |
| | In the past 24 hours, how often were your bowel movements mostly or completely liquid? | 0=Never<br>1=Rarely<br>2=Sometimes<br>3=Often<br>4=Always |
| | In the past 24 hours, did you have blood in your bowel movements? | 0=No<br>1=Rarely<br>2=Sometimes<br>3=Often<br>4=Always |
| | In the past 24 hours, did you have mucus (white material) in your bowel movements? | 0=No<br>1=Rarely<br>2=Sometimes<br>3=Often<br>4=Always |
| | In the past 24 hours, did stool, blood, or liquid leak out before you reached a toilet? | 0=No<br>1=Rarely<br>2=Sometimes<br>3=Often<br>4=Always |
| | In the past 24 hours, did you feel the need to have a bowel movement right away? | 0=No<br>1=Mild<br>2=Moderate<br>3=Severe<br>4=Very Severe |

# Appendix 6 Ulcerative Colitis Patient Reported Outcomes Signs and Symptoms (contd.)

| UC-PRO/SS<br>Domain | Question | Response to<br>Question |
|---|---|---|
| Systemic Symptoms | In the past 24 hours, did you feel pain in your knees, hips, and/or elbows? | 0=No<br>1=Mild<br>2=Moderate<br>3=Severe<br>4=Very Severe |
| | In the past 24 hours, did you feel tired? | 0=No<br>1=Mild<br>2=Moderate<br>3=Severe<br>4=Very Severe |
| | In the past 24 hours, did you lack an appetite? | 0=No<br>1=Mild<br>2=Moderate<br>3=Severe<br>4=Very Severe |
| | In the past 24 hours, did you feel weak? | 0=No<br>1=Mild<br>2=Moderate<br>3=Severe<br>4=Very Severe |
| | In the past 24 hours, did you feel thirsty? | 0=No<br>1=Mild<br>2=Moderate<br>3=Severe<br>4=Very Severe |